CLINICAL TRIAL: NCT02554786
Title: A Multicenter Randomized 52 Week Treatment Double-blind, Triple Dummy Parallel Group Study to Assess the Efficacy and Safety of QMF149 Compared to Mometasone Furoate in Patients With Asthma
Brief Title: A Multicenter Randomized 52 Week Treatment Double-blind, Triple Dummy Parallel Group Study to Assess the Efficacy and Safety of QMF149 Compared to Mometasone Furoate in Participants With Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CQVM149B2301; 2015-002529-21 (EudraCT Number)
Record Dates: First submitted 2015-09-09; First posted 2015-09-18 (Estimated); Results first posted 2020-03-05 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-02

CONDITIONS: Asthma
Keywords: QMF149, Mometasone furoate (MF), asthma
MeSH Terms: conditions — Asthma | interventions — indacaterol; Mometasone Furoate; QMF149; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- QMF149 150/160 µg (Experimental): QMF149 (Indacaterol acetate/Mometasone furoate) 150/160 μg was delivered once daily (o.d) via Concept1 inhaler in the evening.
  Interventions: Drug: Indacaterol acetate/Mometasone furoate
- QMF149 150/320 µg (Experimental): QMF149 (Indacaterol acetate/Mometasone furoate) 150/320 μg was delivered o.d via Concept1 inhaler in the evening.
  Interventions: Drug: Indacaterol acetate/Mometasone furoate
- MF 400 µg (Active Comparator): Mometasone furoate (MF) 400 μg was delivered o.d via Twisthaler® in the evening
  Interventions: Drug: Mometasone furoate
- Salmeterol /fluticasone 50/500 μg (Active Comparator): Salmeterol xinafoate/fluticasone propionate 50/500 μg was delivered twice daily (in the morning and in the evening) via Accuhaler®.
  Interventions: Drug: Salmeterol xinafoate/fluticasone propionate
- MF 800 μg (Active Comparator): MF 800 μg of total daily dose (400 μg twice daily, in the morning and in the evening) was delivered via Twisthaler®.
  Interventions: Drug: Mometasone furoate

INTERVENTIONS:
Drug: Indacaterol acetate/Mometasone furoate
  Other Names: QMF149
  Arms: QMF149 150/160 µg; QMF149 150/320 µg
Drug: Mometasone furoate
  Arms: MF 400 µg; MF 800 μg
Drug: Salmeterol xinafoate/fluticasone propionate
  Arms: Salmeterol /fluticasone 50/500 μg

SUMMARY:
The purpose of the trial is to evaluate the efficacy and safety of two different doses of QMF149 (QMF149 150/160 µg and QMF149 150/320 µg via Concept1) over two respective MF doses (MF 400 µg and MF 800 µg via Twisthaler® (total daily dose)) in poorly controlled asthmatic participants as determined by pulmonary function testing, and effects on asthma control

ELIGIBILITY:
Inclusion Criteria:

* Participants with a diagnosis of asthma, for a period of at least 1 year prior to Visit 1 (Screening)
* Participants who have used medium or high dose inhaled corticosteroids (ICS) or low dose of long acting beta-2 agonist (LABA)/ICS combinations for asthma for at least 3 months and at stable doses for at least 1 month prior to Visit 1
* Participants must have ACQ-7 score ≥ 1.5 at Visit 101 and at Visit 102 (prior to double-blind treatment) and qualify for treatment with medium or high dose LABA/ICS
* Pre-bronchodilator ≥ 50% Forced expiratory volume in 1 second (FEV1) of < 85 % of the predicted normal value for the participants after withholding bronchodilators at both Visit 101 and 102, according to American Thoracic Society/European Respiratory Society (ATS/ERS) criteria.
* Withholding period of bronchodilators prior to spirometry: short acting beta-2 agonist (SABA) for ≥ 6 hours and FDC or free combinations of ICS/LABA for ≥ 48 hours, short acting anticholinergics (SAMA) for ≥ 8 hours, xanthines >=07 days
* A one-time repeat/re-testing of percent predicted FEV1 (prebronchodilator FEV1) is allowed at Visit 101 and at Visit 102.

Spacer devices are permitted for reversibility testing only.

-Participants who demonstrate an increase in FEV1 of 12% and 200 mL within 30 minutes after administration of 400 µg salbutamol/360 µg albuterol (or equivalent dose) at Visit 101 All participants must perform a reversibility test at Visit 101

If reversibility is not demonstrated at Visit 101:

* Reversibility should be repeated once-
* Participants may be permitted to enter the study with historical evidence of reversibility that was performed according to ATS/ERS guidelines within 2 years prior to Visit 1
* Alternatively, participants may be permitted to enter the study with a historical positive bronchoprovocation test that was performed within 2 years prior to Visit 1.

Exclusion Criteria:

* Participants who have smoked or inhaled tobacco products within the 6 month period prior to Visit 1, or who have a smoking history of greater than 10 pack years. This includes use of nicotine inhalers such as e-cigarettes at the time of Visit 1
* Participants who have had an asthma attack/exacerbation requiring systemic steroids or hospitalization or emergency room visit within 6 weeks of Visit 1 (Screening)
* Participants who have ever required intubation for a severe asthma attack/exacerbation.
* Participants who have a clinical condition which is likely to be worsened by ICS administration (e.g. glaucoma, cataract and fragility fractures) who are according to investigator's medical judgment at risk participating in the study).
* Participants who have had a respiratory tract infection or asthma worsening as determined by the investigator within 4 weeks prior to Visit 1 (Screening) or between Visit 1 and Visit 102. Participants may be re-screened 4 weeks after recovery from their respiratory tract infection or asthma worsening.
* Participants with a history of chronic lung diseases other than asthma, including (but not limited to) Chronic Obstructive Pulmonary Disease (COPD), sarcoidosis, interstitial lung disease, cystic fibrosis, clinically significant bronchiectasis and active tuberculosis.
* Participants with severe narcolepsy and/or insomnia.
* Participants who have a clinically significant electrocardiogram (ECG) abnormality at Visit 101 (Start of Run- In epoch) and at any time between Visit 101 and Visit 102 (including unscheduled ECG). ECG evidence of myocardial infarction at Visit 101 (via central reader) should be clinically assessed by the investigator with supportivedocumentation
* Participants with a history of hypersensitivity to lactose, any of the study drugs or to similar drugs within the class including untoward reactions to sympathomimetic amines or inhaled medication or any component thereof
* Participants who have not achieved an acceptable spirometry results at Visit 101 in accordance with ATS/ERS criteria for acceptability and repeatability (rescreening allowed only once).

Repeat spirometry may be allowed once in an ad-hoc visit if the spirometry did not qualify due to ATS/ERS criteria. If the participant fails the repeat assessment, the participant may be rescreened once

* Participants on Maintenance Immunotherapy (desensitization) for allergies or less than 3 months prior to Visit 101 or participants on Maintenance Immunotherapy for more than 3 months prior to Visit 101 but expected to change throughout the course of the study.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing of study treatment and for 30 days after stopping of study treatment.
* Long acting muscarinic antagonist (LAMA) use within 3 months prior to Visit 101

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2216 (Actual)
Dates: Start 2015-12-29 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2019-06-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (306):
- United States (29):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Orange, California
  - Novartis Investigative Site, Riverside, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, San Jose, California
  - Novartis Investigative Site, Stockton, California
  - Novartis Investigative Site, Westminster, California
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Tallahassee, Florida
  - Novartis Investigative Site, Winter Park, Florida
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Waldorf, Maryland
  - Novartis Investigative Site, North Dartmouth, Massachusetts
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Bellevue, Nebraska
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Skillman, New Jersey
  - Novartis Investigative Site, Cortland, New York
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Tulsa, Oklahoma
  - Novartis Investigative Site, Medford, Oregon
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, North Charleston, South Carolina
  - Novartis Investigative Site, Boerne, Texas
  - Novartis Investigative Site, El Paso, Texas
  - Novartis Investigative Site, Greenfield, Wisconsin
- Bulgaria (9):
  - Novartis Investigative Site, Plovdiv, BGR
  - Novartis Investigative Site, Varna, BGR
  - Novartis Investigative Site, Vidin, BGR
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Rousse
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Stara Zagora
  - Novartis Investigative Site, Troyan Municipality
- China (22):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Fuzhou, Fujian
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Haikou, Hainan
  - Novartis Investigative Site, Shijiazhuang, Hebei
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Suzhou, Jiangsu
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Shanghai, Shanghai Municipality
  - Novartis Investigative Site, Xian, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Chengdu
  - Novartis Investigative Site, Chongqing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Nanchang
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- Croatia (6):
  - Novartis Investigative Site, Varaždin, HRV
  - Novartis Investigative Site, Zagreb, HRV
  - Novartis Investigative Site, Petrinja
  - Novartis Investigative Site, Rijeka
  - Novartis Investigative Site, Zadar
  - Novartis Investigative Site, Zagreb
- Czechia (19):
  - Novartis Investigative Site, Beroun, Czech Republic
  - Novartis Investigative Site, Boskovice, Czech Republic
  - Novartis Investigative Site, Jablonec nad Nisou, Czech Republic
  - Novartis Investigative Site, Jindřichův Hradec, Czech Republic
  - Novartis Investigative Site, Kuřim, Czech Republic
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Teplice, Czech Republic
  - Novartis Investigative Site, Varnsdorf, Czech Republic
  - Novartis Investigative Site, Ostrava, CZE
  - Novartis Investigative Site, Pilsen, CZE
  - Novartis Investigative Site, Teplice, CZE
  - Novartis Investigative Site, Břeclav
  - Novartis Investigative Site, Český Krumlov
  - Novartis Investigative Site, Kutná Hora
  - Novartis Investigative Site, Nový Bor
  - Novartis Investigative Site, Pilsen
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Rokycany
  - Novartis Investigative Site, Tábor
- Novartis Investigative Site, Alexandria, Egypt
- Estonia (2):
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- Germany (35):
  - Novartis Investigative Site, Peine, Lower Saxony
  - Novartis Investigative Site, Koblenz, Rhineland-Palatinate
  - Novartis Investigative Site, Ahlen
  - Novartis Investigative Site, Bamberg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Böhlen
  - Novartis Investigative Site, Delitzsch
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Düren
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Fürstenwalde
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Hochstadt
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Ludwigsburg
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Mittweida
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Neu-Isenburg
  - Novartis Investigative Site, Neuss
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Rheine
  - Novartis Investigative Site, Rüdersdorf
  - Novartis Investigative Site, Schleswig
  - Novartis Investigative Site, Schwedt
  - Novartis Investigative Site, Weinheim
  - Novartis Investigative Site, Witten
- Guatemala (3):
  - Novartis Investigative Site, Ciudad, Gautemala
  - Novartis Investigative Site, Guatemala City, GTM
  - Novartis Investigative Site, Guatemala City
- Hungary (21):
  - Novartis Investigative Site, Budapest, HUN
  - Novartis Investigative Site, Győr, HUN
  - Novartis Investigative Site, Hajdúnánás, HUN
  - Novartis Investigative Site, Makó, HUN
  - Novartis Investigative Site, Miskolc, HUN
  - Novartis Investigative Site, Püspökladány, HUN
  - Novartis Investigative Site, Százhalombatta, HUN
  - Novartis Investigative Site, Balassagyarmat
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Cegléd
  - Novartis Investigative Site, Csorna
  - Novartis Investigative Site, Dombóvár
  - Novartis Investigative Site, Gödöllő
  - Novartis Investigative Site, Hatvan
  - Novartis Investigative Site, Komárom
  - Novartis Investigative Site, Miskolc
  - Novartis Investigative Site, Mosdós
  - Novartis Investigative Site, Szarvas
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Szigetvár
  - Novartis Investigative Site, Szombathely
- India (13):
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Vadodara, Gujarat
  - Novartis Investigative Site, Mysore, Karnataka
  - Novartis Investigative Site, Kozhikode, Kerala
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Mohali, Punjab
  - Novartis Investigative Site, Jaipur, Rajasthan
  - Novartis Investigative Site, Hyderabad, Telangana
  - Novartis Investigative Site, Lucknow, Uttar Pradesh
  - Novartis Investigative Site, New Delhi
- Ireland (3):
  - Novartis Investigative Site, Wilton, Cork
  - Novartis Investigative Site, County Limerick
  - Novartis Investigative Site, Dublin
- Japan (26):
  - Novartis Investigative Site, Ichihara, Chiba
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kasuga, Fukuoka
  - Novartis Investigative Site, Yanagawa, Fukuoka
  - Novartis Investigative Site, Obihiro, Hokkaido
  - Novartis Investigative Site, Himeji, Hyōgo
  - Novartis Investigative Site, Naka-gun, Ibaraki
  - Novartis Investigative Site, Atsugi, Kanagawa
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Okayama, Okayama-ken
  - Novartis Investigative Site, Kishiwada, Osaka
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Takatsuki, Osaka
  - Novartis Investigative Site, Toyonaka, Osaka
  - Novartis Investigative Site, Yao, Osaka
  - Novartis Investigative Site, Koshigaya, Saitama
  - Novartis Investigative Site, Tokyo, Shibuya Ku
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Chuou-ku, Tokyo
  - Novartis Investigative Site, Itabashi-ku, Tokyo
  - Novartis Investigative Site, Setagaya-Ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Toshima Ku, Tokyo
  - Novartis Investigative Site, Toshima-ku, Tokyo
- Latvia (3):
  - Novartis Investigative Site, Riga, LV
  - Novartis Investigative Site, Daugavpils
  - Novartis Investigative Site, Riga
- Lithuania (5):
  - Novartis Investigative Site, Kaunas, LTU
  - Novartis Investigative Site, Kaunas
  - Novartis Investigative Site, Šiauliai
  - Novartis Investigative Site, Utena
  - Novartis Investigative Site, Vilnius
- Mexico (3):
  - Novartis Investigative Site, Mexicali, Estado de Baja California
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, México
- Poland (14):
  - Novartis Investigative Site, Aleksandrow Odzki, Poland
  - Novartis Investigative Site, Biaystok, Poland
  - Novartis Investigative Site, Lodz, POL
  - Novartis Investigative Site, Wejherowo, POL
  - Novartis Investigative Site, Bielsko-Biala
  - Novartis Investigative Site, Elblag
  - Novartis Investigative Site, Inowrocław
  - Novartis Investigative Site, Katowice
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Ostrów Wielkopolski
  - Novartis Investigative Site, Sopot
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Zawadzkie
- Romania (20):
  - Novartis Investigative Site, Iași, Jud Iasi
  - Novartis Investigative Site, Constanța, Jud. Constanta
  - Novartis Investigative Site, Craiova, Jud.Dolj
  - Novartis Investigative Site, Bucharest, ROM
  - Novartis Investigative Site, Craiova, ROM
  - Novartis Investigative Site, Deva, ROM
  - Novartis Investigative Site, Timișoara, ROM
  - Novartis Investigative Site, Timișoara, Timiș County
  - Novartis Investigative Site, Arad
  - Novartis Investigative Site, Bacau
  - Novartis Investigative Site, Bragadiru
  - Novartis Investigative Site, Brasov
  - Novartis Investigative Site, Brăila
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Cluj-Napoca
  - Novartis Investigative Site, Codlea
  - Novartis Investigative Site, Craiova
  - Novartis Investigative Site, Râmnicu Vâlcea
  - Novartis Investigative Site, Suceava
  - Novartis Investigative Site, Târgu Mureş
- Russia (19):
  - Novartis Investigative Site, Yaroslavl, Russian Federation
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Krasnoyarsk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, N.Novgorod
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, Penza
  - Novartis Investigative Site, Petrozavodsk
  - Novartis Investigative Site, Pyatigorsk
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Saratov
  - Novartis Investigative Site, Smolensk
  - Novartis Investigative Site, Stavropol
  - Novartis Investigative Site, Volgograd
  - Novartis Investigative Site, Vologodonsk
  - Novartis Investigative Site, Yaroslavl
  - Novartis Investigative Site, Yekaterinburg
- Serbia (5):
  - Novartis Investigative Site, Belgrade, Serbia
  - Novartis Investigative Site, Belgrade
  - Novartis Investigative Site, Kamenitz
  - Novartis Investigative Site, Kragujevac
  - Novartis Investigative Site, Niš
- Slovakia (26):
  - Novartis Investigative Site, Bardejov, Slovak Republic
  - Novartis Investigative Site, Bojnice, Slovak Republic
  - Novartis Investigative Site, Bratislava, Slovak Republic
  - Novartis Investigative Site, Humenné, Slovak Republic
  - Novartis Investigative Site, Košice, Slovak Republic
  - Novartis Investigative Site, Nitra, Slovak Republic
  - Novartis Investigative Site, Skalica, Slovak Republic
  - Novartis Investigative Site, Spišská Nová Ves, Slovak Republic
  - Novartis Investigative Site, Stropkov, Slovak Republic
  - Novartis Investigative Site, Šurany, Slovak Republic
  - Novartis Investigative Site, Veľký Meder, Slovak Republic
  - Novartis Investigative Site, Námestovo, Slovensko
  - Novartis Investigative Site, Poprad, SVK
  - Novartis Investigative Site, Bardejov
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Čadca
  - Novartis Investigative Site, Ilava
  - Novartis Investigative Site, Komárno
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Kráľovský Chlmec
  - Novartis Investigative Site, Levice
  - Novartis Investigative Site, Liptovský Mikuláš
  - Novartis Investigative Site, Prešov
  - Novartis Investigative Site, Prievidza
  - Novartis Investigative Site, Topoľčany
  - Novartis Investigative Site, Žilina
- South Africa (4):
  - Novartis Investigative Site, Berea, Durban
  - Novartis Investigative Site, Belleville, South Africa
  - Novartis Investigative Site, Panorama, Western Cape
  - Novartis Investigative Site, Cape Town
- South Korea (7):
  - Novartis Investigative Site, Wŏnju, Gangwon-do
  - Novartis Investigative Site, Bucheon-si, Gyeonggi-do
  - Novartis Investigative Site, Bundang Gu, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Cheongju-si, North Chungcheong
  - Novartis Investigative Site, Seoul, Seocho Gu
  - Novartis Investigative Site, Incheon
- United Kingdom (11):
  - Novartis Investigative Site, Fowey, Cornwall
  - Novartis Investigative Site, Liskeard, Cornwall
  - Novartis Investigative Site, Torpoint, Cornwall
  - Novartis Investigative Site, Faringdon, Oxfordshire
  - Novartis Investigative Site, Bristol, South Gloucestershire
  - Novartis Investigative Site, Blackpool
  - Novartis Investigative Site, Denbighshire
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Rotherham
  - Novartis Investigative Site, Wiltshire

REFERENCES:
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162
- [Derived] Chapman K, van Zyl-Smit R, Maspero J, Kerstjens HAM, Gon Y, Hosoe M, Tanase AM, Pethe A, Shu X, D'Andrea P. One time a day mometasone/indacaterol fixed-dose combination versus two times a day fluticasone/salmeterol in patients with inadequately controlled asthma: pooled analysis from PALLADIUM and IRIDIUM studies. BMJ Open Respir Res. 2021 Aug;8(1):e000819. doi: 10.1136/bmjresp-2020-000819. PMID 34452934
- [Derived] van Zyl-Smit RN, Krull M, Gessner C, Gon Y, Noga O, Richard A, de Los Reyes A, Shu X, Pethe A, Tanase AM, D'Andrea P; PALLADIUM trial investigators. Once-daily mometasone plus indacaterol versus mometasone or twice-daily fluticasone plus salmeterol in patients with inadequately controlled asthma (PALLADIUM): a randomised, double-blind, triple-dummy, controlled phase 3 study. Lancet Respir Med. 2020 Oct;8(10):987-999. doi: 10.1016/S2213-2600(20)30178-8. Epub 2020 Jul 9. PMID 32653075

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 316 investigative sites in 24 countries from 29 Dec 2015 to 28 Jun 2019.
Pre-assignment Details: 3890 participants were screened of which 2216 were randomized to 1 of the 5 treatment groups with a randomization ratio of 1:1:1:1:1.
Groups:
- QMF149 150/320 μg: QMF149 (Indacaterol acetate/Mometasone furoate) 150/320 μg was delivered once daily (o.d.) via Concept1 inhaler in the evening.
- QMF149 150/160 μg: QMF149 (Indacaterol acetate/Mometasone furoate) 150/160 μg was delivered o.d. via Concept1 inhaler in the evening.
- MF 800 μg: Mometasone furoate (MF) 800 μg of total daily dose (400 μg twice daily, in the morning and in the evening) was delivered via Twisthaler®.
- MF 400 μg: MF 400 μg was delivered o.d. via Twisthaler® in the evening.
- Salmeterol/Fluticasone 50/500 μg: Salmeterol xinafoate/fluticasone propionate 50/500 μg was delivered twice daily (in the morning and in the evening) via Accuhaler®.
Period: Overall Study
Arm/Group | QMF149 150/320 μg | QMF149 150/160 μg | MF 800 μg | MF 400 μg | Salmeterol/Fluticasone 50/500 μg
Started | 445 | 439 | 442 | 444 | 446
Completed | 410 | 413 | 412 | 403 | 416
Not Completed | 35 | 26 | 30 | 41 | 30
Not completed — Subject/guardian decision | 29 | 17 | 18 | 30 | 20
Not completed — Lost to Follow-up | 4 | 3 | 4 | 2 | 2
Not completed — Protocol deviation | 1 | 3 | 3 | 4 | 2
Not completed — Technical problems | 1 | 1 | 0 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2
Not completed — Death | 0 | 0 | 0 | 1 | 0
Not completed — Non-compliance with study treatment | 0 | 1 | 1 | 0 | 1
Not completed — Physician Decision | 0 | 1 | 4 | 1 | 1
Not completed — Pregnancy | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Randomized Set (RAN) consisted of all participants who were assigned a randomization number, regardless of whether or not they actually received study medication.
Groups:
- QMF149 150/320 μg: QMF149 (Indacaterol acetate/Mometasone furoate) 150/320 μg was delivered o.d. via Concept1 inhaler in the evening.
- Total: Total of all reporting groups
Arm/Group | QMF149 150/320 μg | QMF149 150/160 μg | MF 800 μg | MF 400 μg | Salmeterol/Fluticasone 50/500 μg | Total
Number analyzed (Participants) | 445 | 439 | 442 | 444 | 446 | 2216
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (14.56) | 47.4 (14.76) | 47.5 (14.99) | 48.7 (14.98) | 48.9 (14.59) | 47.9 (14.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 262 | 253 | 250 | 272 | 256 | 1293
  Male | 183 | 186 | 192 | 172 | 190 | 923
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 313 | 311 | 318 | 312 | 305 | 1559
  Race: Black | 5 | 2 | 4 | 8 | 4 | 23
  Race: Asian | 97 | 98 | 98 | 98 | 102 | 493
  Race: Native American | 13 | 14 | 11 | 18 | 12 | 68
  Race: Pacific Islander | 1 | 0 | 0 | 0 | 0 | 1
  Race: Other | 16 | 14 | 11 | 8 | 23 | 72
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic Or Latino | 21 | 17 | 14 | 22 | 15 | 89
  Ethnicity: East Asian | 52 | 48 | 51 | 55 | 53 | 259
  Ethnicity: Southeast Asian | 38 | 40 | 42 | 38 | 42 | 200
  Ethnicity: South Asian | 3 | 3 | 2 | 3 | 3 | 14
  Ethnicity: Russian | 79 | 79 | 64 | 62 | 65 | 349
  Ethnicity: Mixed ethnicity | 10 | 10 | 9 | 5 | 15 | 49
  Ethnicity: Not reported | 12 | 4 | 12 | 5 | 9 | 42
  Ethnicity: Unknown | 12 | 13 | 6 | 15 | 17 | 63
  Ethnicity: Other | 218 | 225 | 242 | 239 | 227 | 1151

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratory Volume in One Second (Trough FEV1) at Week 26
Description: Trough FEV1 was assessed by performing spirometric assessment. It is defined as average of the two FEV1 measurements taken 23 hr 15 min and 23 hr 45 min post-evening dose. FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation, measured through spirometry testing.
Time Frame: 26 weeks
Population: Full Analysis Set (FAS) consisted of all participants in the RAN set who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: litre (L)
Arm/Group | QMF149 150/320 μg | QMF149 150/160 μg | MF 800 μg | MF 400 μg | Salmeterol/Fluticasone 50/500 μg
Number analyzed (Participants) | 395 | 389 | 372 | 376 | 391
litre (L) | 2.383 (0.0159) | 2.387 (0.0160) | 2.250 (0.0162) | 2.176 (0.0162) | 2.346 (0.0160)
Statistical Analysis 1: Comparison: QMF149 150/320 μg vs MF 800 μg; Test type: Superiority; p < 0.001, Mixed Model for Repeated Measures (MMRM); Least Square mean (LS Mean) = 0.132, 95% CI 2-sided [0.088 to 0.176], Standard Error of Mean 0.0223
Statistical Analysis 2: Comparison: QMF149 150/160 μg vs MF 400 μg; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.211, 95% CI 2-sided [0.167 to 0.255], Standard Error of Mean 0.0224

2. Secondary Outcome: Asthma Control Questionnaire (ACQ-7) at Weeks 4, 12, 26 and 52
Description: The ACQ-7 measured asthma symptom control and consists of 7 items: 5 on symptom assessment, 1 on rescue bronchodilator use and 1 on airway calibre (FEV1 % predicted). All 7 questions of the ACQ-7 were equally weighted. Items 1-5 were scored along a 7-point response scale, where 0 = totally controlled and 6 = severely uncontrolled. Item 6 is scored between 0 = no rescue medication and 6 = More than 16 puffs/inhalations most days. The 7th item was scored by the investigator based on the FEV1 % predicted from the masterscope at the site (i.e., Score = 0 means > 95% of predicted FEV1, 1 = 90 - 95%, 2 = 80 - 89%, 3 = 70 - 79%, 4 = 60 - 69%, 5 = 50 - 59%, and Score = 6 means < 50% of predicted FEV1). The total score was calculated as the mean of all questions.
Time Frame: Weeks 4, 12, 26 and 52
Population: FAS consisted of all participants in the RAN set who received at least one dose of study medication. n represents the number of participants with data at respective visit
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | QMF149 150/320 μg | QMF149 150/160 μg | MF 800 μg | MF 400 μg | Salmeterol/Fluticasone 50/500 μg
Number analyzed (Participants) | 429 | 427 | 431 | 428 | 439
score on a scale
  Week 4: number analyzed (Participants) | 426 | 422 | 429 | 425 | 437
  Week 4 | 1.486 (0.0337) | 1.533 (0.0338) | 1.659 (0.0338) | 1.730 (0.0337) | 1.541 (0.0335)
  Week 12: number analyzed (Participants) | 419 | 414 | 422 | 407 | 429
  Week 12 | 1.394 (0.0347) | 1.377 (0.0348) | 1.523 (0.0348) | 1.625 (0.0350) | 1.445 (0.0345)
  Week 26: number analyzed (Participants) | 407 | 407 | 405 | 393 | 410
  Week 26 | 1.267 (0.0350) | 1.261 (0.0350) | 1.439 (0.0352) | 1.509 (0.0354) | 1.322 (0.0349)
  Week 52: number analyzed (Participants) | 385 | 397 | 387 | 377 | 405
  Week 52 | 1.231 (0.0358) | 1.183 (0.0356) | 1.373 (0.0359) | 1.449 (0.0361) | 1.221 (0.0354)
Statistical Analysis 1: Comparison: QMF149 150/320 μg vs MF 800 μg; Week 4; Test type: Superiority; p < 0.001, MMRM; LS Mean = -0.172, 95% CI 2-sided [-0.254 to -0.091], Standard Error of Mean 0.0415
Statistical Analysis 2: Comparison: QMF149 150/160 μg vs MF 400 μg; Week 4; Test type: Superiority; p < 0.001, MMRM; LS Mean = -0.196, 95% CI 2-sided [-0.278 to -0.115], Standard Error of Mean 0.0416
Statistical Analysis 3: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Week 4; Test type: Superiority; p = 0.186, MMRM; LS Mean = -0.055, 95% CI 2-sided [-0.136 to 0.026], Standard Error of Mean 0.0414
Statistical Analysis 4: Comparison: QMF149 150/320 μg vs QMF149 150/160 μg vs MF 800 μg vs MF 400 μg; Week 4: The comparison of QMF149 vs. MF was based on combined effects of QMF149 150/160 & 150/320 μg and MF 400 & 800 μg derived by weighting treatment groups equally; Test type: Superiority; p < 0.001, MMRM; LS Mean = -0.184, 95% CI 2-sided [-0.242 to -0.127], Standard Error of Mean 0.0294
Statistical Analysis 5: Comparison: QMF149 150/320 μg vs MF 800 μg; Week 12; Test type: Superiority; p = 0.003, MMRM; LS Mean = -0.129, 95% CI 2-sided [-0.214 to -0.044], Standard Error of Mean 0.0431
Statistical Analysis 6: Comparison: QMF149 150/160 μg vs MF 400 μg; Week 12; Test type: Superiority; p < 0.001, MMRM; LS Mean = -0.248, 95% CI 2-sided [-0.333 to -0.162], Standard Error of Mean 0.0435
Statistical Analysis 7: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Week 12; Test type: Superiority; p = 0.232, MMRM; LS Mean = -0.052, 95% CI 2-sided [-0.136 to 0.033], Standard Error of Mean 0.0431
Statistical Analysis 8: Comparison: QMF149 150/320 μg vs QMF149 150/160 μg vs MF 800 μg vs MF 400 μg; Week 12: The comparison of QMF149 vs. MF was based on combined effects of QMF149 150/160 & 150/320 μg and MF 400 & 800 μg derived by weighting treatment groups equally; Test type: Superiority; p < 0.001, MMRM; LS Mean = -0.188, 95% CI 2-sided [-0.248 to -0.128], Standard Error of Mean 0.0307
Statistical Analysis 9: Comparison: QMF149 150/320 μg vs MF 800 μg; Week 26; Test type: Superiority; p < 0.001, MMRM; LS Mean = -0.171, 95% CI 2-sided [-0.257 to -0.086], Standard Error of Mean 0.0437
Statistical Analysis 10: Comparison: QMF149 150/160 μg vs MF 400 μg; Week 26; Test type: Superiority; p < 0.001, MMRM; LS Mean = -0.248, 95% CI 2-sided [-0.334 to -0.162], Standard Error of Mean 0.0439
Statistical Analysis 11: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Week 26; Test type: Superiority; p = 0.214, MMRM; LS Mean = -0.054, 95% CI 2-sided [-0.140 to 0.031], Standard Error of Mean 0.0437
Statistical Analysis 12: Comparison: QMF149 150/320 μg vs QMF149 150/160 μg vs MF 800 μg vs MF 400 μg; Week 26: The comparison of QMF149 vs. MF was based on combined effects of QMF149 150/160 & 150/320 μg and MF 400 & 800 μg derived by weighting treatment groups equally; Test type: Superiority; p < 0.001, MMRM; LS Mean = -0.209, 95% CI 2-sided [-0.270 to -0.149], Standard Error of Mean 0.0310
Statistical Analysis 13: Comparison: QMF149 150/320 μg vs MF 800 μg; Week 52; Test type: Superiority; p = 0.002, MMRM; LS Mean = -0.141, 95% CI 2-sided [-0.229 to -0.053], Standard Error of Mean 0.0449
Statistical Analysis 14: Comparison: QMF149 150/160 μg vs MF 400 μg; Week 52; Test type: Superiority; p < 0.001, MMRM; LS Mean = -0.266, 95% CI 2-sided [-0.354 to -0.177], Standard Error of Mean 0.045
Statistical Analysis 15: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Week 52; Test type: Superiority; p = 0.824, MMRM; LS Mean = 0.01, 95% CI 2-sided [-0.078 to 0.098], Standard Error of Mean 0.0447
Statistical Analysis 16: Comparison: QMF149 150/320 μg vs QMF149 150/160 μg vs MF 800 μg vs MF 400 μg; Week 52: The comparison of QMF149 vs. MF was based on combined effects of QMF149 150/160 & 150/320 μg and MF 400 & 800 μg derived by weighting treatment groups equally; Test type: Superiority; p < 0.001, MMRM; LS Mean = -0.203, 95% CI 2-sided [-0.266 to -0.141], Standard Error of Mean 0.0318

3. Secondary Outcome: Trough FEV1 at Week 52
Description: as for outcome 1
Time Frame: Week 52
Population: FAS consisted of all participants in the RAN set who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | QMF149 150/320 μg | QMF149 150/160 μg | MF 800 μg | MF 400 μg | Salmeterol/Fluticasone 50/500 μg
Number analyzed (Participants) | 372 | 383 | 364 | 369 | 382
L | 2.386 (0.0168) | 2.357 (0.0167) | 2.249 (0.0170) | 2.148 (0.0170) | 2.338 (0.0167)
Statistical Analysis 1: Comparison: QMF149 150/320 μg vs MF 800 μg; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.136, 95% CI 2-sided [0.090 to 0.183], Standard Error of Mean 0.0235
Statistical Analysis 2: Comparison: QMF149 150/160 μg vs MF 400 μg; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.209, 95% CI 2-sided [0.163 to 0.255], Standard Error of Mean 0.0235
Statistical Analysis 3: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Test type: Superiority; p = 0.04, MMRM; LS Mean = 0.048, 95% CI 2-sided [0.002 to 0.094], Standard Error of Mean 0.0234

4. Secondary Outcome: Pre-dose FEV1 at Weeks 4 and 12
Description: Pre-dose trough FEV1 is defined as average of the two FEV1 measurements taken 45 min and 15 min pre evening dose. It was assessed by performing spirometric assessment. FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation, measured through spirometry testing.
Time Frame: Weeks 4 (Day 30) and 12 (Day 86)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Deviation); unit: L
Groups:
- MF 400 μg: MF 400 μg was delivered o.d via Twisthaler® in the evening
Arm/Group | QMF149 150/320 μg | QMF149 150/160 μg | MF 800 μg | MF 400 μg | Salmeterol /Fluticasone 50/500 μg
Number analyzed (Participants) | 430 | 427 | 430 | 427 | 439
L
  Day 30: number analyzed (Participants) | 430 | 424 | 421 | 412 | 435
  Day 30 | 2.369 (0.0141) | 2.367 (0.0142) | 2.237 (0.0143) | 2.171 (0.0143) | 0.2333 (0.0141)
  Day 86: number analyzed (Participants) | 414 | 414 | 419 | 398 | 428
  Day 86 | 2.368 (0.0148) | 2.361 (0.0148) | 2.245 (0.0148) | 2.177 (0.0149) | 2.330 (0.0146)
Statistical Analysis 1: Comparison: QMF149 150/320 μg vs MF 800 μg; Day 30; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.132, 95% CI 2-sided [0.094 to 0.170], Standard Error of Mean 0.0193
Statistical Analysis 2: Comparison: QMF149 150/160 μg vs MF 400 μg; Day 30; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.196, 95% CI 2-sided [0.158 to 0.234], Standard Error of Mean 0.0194
Statistical Analysis 3: Comparison: QMF149 150/320 μg vs Salmeterol /Fluticasone 50/500 μg; Day 30; Test type: Superiority; p = 0.064, MMRM; LS Mean = 0.035, 95% CI 2-sided [-0.002 to 0.073], Standard Error of Mean 0.0192
Statistical Analysis 4: Comparison: QMF149 150/320 μg vs MF 800 μg; Day 86; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.122, 95% CI 2-sided [0.083 to 0.162], Standard Error of Mean 0.0201
Statistical Analysis 5: Comparison: QMF149 150/160 μg vs MF 400 μg; Day 86; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.184, 95% CI 2-sided [0.144 to 0.224], Standard Error of Mean 0.0202
Statistical Analysis 6: Comparison: QMF149 150/320 μg vs Salmeterol /Fluticasone 50/500 μg; Day 86; Test type: Superiority; p = 0.063, MMRM; LS Mean = 0.037, 95% CI 2-sided [-0.002 to 0.076], Standard Error of Mean 0.02

5. Secondary Outcome: Post Dose FEV1 (5 Minutes-1 Hour)
Description: Post-dose FEV1 measurements were analyzed at 5 minutes, 15 minutes, 30 minutes and 1 hour. FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation, measured through spirometry testing.
Time Frame: Up to Week 52 (Day 364)
Population: FAS consisted of all participants in the RAN set who received at least one dose of study medication. n represents the number of participants with data at respective time point.
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | QMF149 150/320 μg | QMF149 150/160 μg | MF 800 μg | MF 400 μg | Salmeterol/Fluticasone 50/500 μg
Number analyzed (Participants) | 441 | 434 | 438 | 438 | 442
L
  Day 1: 5 minutes: number analyzed (Participants) | 427 | 426 | 429 | 432 | 435
  Day 1: 5 minutes | 2.279 (0.0084) | 2.270 (0.0085) | 2.138 (0.0085) | 2.118 (0.0084) | 2.224 (0.0084)
  Day 1: 15 minutes: number analyzed (Participants) | 434 | 425 | 433 | 433 | 441
  Day 1: 15 minutes | 2.321 (0.0088) | 2.312 (0.0089) | 2.159 (0.0089) | 2.137 (0.0089) | 2.278 (0.0088)
  Day 1: 30 minutes: number analyzed (Participants) | 439 | 431 | 434 | 438 | 441
  Day 1: 30 minutes | 2.338 (0.0095) | 2.326 (0.0096) | 2.162 (0.0096) | 2.141 (0.0095) | 2.310 (0.0095)
  Day 1: 1 hour: number analyzed (Participants) | 440 | 434 | 435 | 438 | 442
  Day 1: 1 hour | 2.343 (0.0100) | 2.347 (0.0101) | 2.166 (0.0101) | 2.142 (0.0100) | 2.337 (0.0100)
  Day 30: 5 minutes: number analyzed (Participants) | 428 | 420 | 419 | 411 | 435
  Day 30: 5 minutes | 2.413 (0.0142) | 2.406 (0.0144) | 2.224 (0.0145) | 2.174 (0.0145) | 2.360 (0.0142)
  Day 30: 30 minutes: number analyzed (Participants) | 429 | 420 | 421 | 412 | 435
  Day 30: 30 minutes | 2.432 (0.0143) | 2.426 (0.0145) | 2.238 (0.0146) | 2.174 (0.0146) | 2.389 (0.0143)
  Day 30: 1 hour: number analyzed (Participants) | 428 | 416 | 421 | 410 | 435
  Day 30: 1 hour | 2.448 (0.0145) | 2.440 (0.0146) | 2.257 (0.0147) | 2.183 (0.0148) | 2.411 (0.0144)
  Day 86:5 minutes: number analyzed (Participants) | 411 | 411 | 416 | 395 | 427
  Day 86:5 minutes | 2.411 (0.0150) | 2.409 (0.0150) | 2.248 (0.0150) | 2.178 (0.0153) | 2.356 (0.0148)
  Day 86: 30 minutes: number analyzed (Participants) | 412 | 411 | 417 | 395 | 426
  Day 86: 30 minutes | 2.436 (0.0149) | 2.431 (0.0149) | 2.257 (0.0149) | 2.179 (0.0152) | 2.398 (0.0147)
  Day 86:1 hour: number analyzed (Participants) | 412 | 410 | 417 | 396 | 426
  Day 86:1 hour | 2.456 (0.0151) | 2.436 (0.0151) | 2.269 (0.0151) | 2.188 (0.0154) | 2.413 (0.0149)
  Day 183: 5 minutes: number analyzed (Participants) | 404 | 399 | 400 | 385 | 409
  Day 183: 5 minutes | 2.403 (0.0160) | 2.406 (0.0161) | 2.240 (0.0162) | 2.163 (0.0164) | 2.359 (0.0160)
  Day 183: 30 minutes: number analyzed (Participants) | 405 | 401 | 399 | 383 | 407
  Day 183: 30 minutes | 2.426 (0.0163) | 2.427 (0.0164) | 2.250 (0.0165) | 2.168 (0.0167) | 2.386 (0.0163)
  Day 183: 1 hour: number analyzed (Participants) | 405 | 400 | 397 | 385 | 409
  Day 183: 1 hour | 2.432 (0.0161) | 2.423 (0.0162) | 2.253 (0.0163) | 2.165 (0.0165) | 2.393 (0.0161)
  Day 364: 5 minutes: number analyzed (Participants) | 375 | 389 | 380 | 374 | 403
  Day 364: 5 minutes | 2.384 (0.0172) | 2.379 (0.0169) | 2.245 (0.0172) | 2.130 (0.0173) | 2.358 (0.0168)
  Day 364: 30 minutes: number analyzed (Participants) | 377 | 393 | 379 | 373 | 401
  Day 364: 30 minutes | 2.408 (0.0171) | 2.399 (0.0169) | 2.253 (0.0172) | 2.135 (0.0172) | 2.377 (0.0167)
  Day 364:1 hour: number analyzed (Participants) | 378 | 393 | 379 | 375 | 402
  Day 364:1 hour | 2.414 (0.0175) | 2.390 (0.0172) | 2.251 (0.0175) | 2.128 (0.0176) | 2.383 (0.0171)
Statistical Analysis 1: Comparison: QMF149 150/320 μg vs MF 800 μg; Day 1: 5 minutes; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.142, 95% CI 2-sided [0.119 to 0.164], Standard Error of Mean 0.0116
Statistical Analysis 2: Comparison: QMF149 150/160 μg vs MF 400 μg; Day 1: 5 minutes; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.152, 95% CI 2-sided [0.129 to 0.175], Standard Error of Mean 0.0116
Statistical Analysis 3: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Day 1: 5 minutes; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.055, 95% CI 2-sided [0.032 to 0.078], Standard Error of Mean 0.0116
Statistical Analysis 4: Comparison: QMF149 150/320 μg vs MF 800 μg; Day 1: 15 minutes; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.162, 95% CI 2-sided [0.138 to 0.186], Standard Error of Mean 0.0122
Statistical Analysis 5: Comparison: QMF149 150/160 μg vs MF 400 μg; Day 1: 15 minutes; Test type: Superiority; p < .001, MMRM; LS mean = 0.174, 95% CI 2-sided [0.150 to 0.198], Standard Error of Mean 0.0123
Statistical Analysis 6: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Day1: 15 minutes; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.044, 95% CI 2-sided [0.02 to 0.068], Standard Error of Mean 0.0122
Statistical Analysis 7: Comparison: QMF149 150/320 μg vs MF 800 μg; Day 1: 30 minutes; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.175, 95% CI 2-sided [0.149 to 0.201], Standard Error of Mean 0.0132
Statistical Analysis 8: Comparison: QMF149 150/160 μg vs MF 400 μg; Day 1: 30 minutes; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.185, 95% CI 2-sided [0.159 to 0.211], Standard Error of Mean 0.0132
Statistical Analysis 9: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Day 1: 30 minutes; Test type: Superiority; p = 0.038, MMRM; LS Mean = 0.027, 95% CI 2-sided [0.001 to 0.053], Standard Error of Mean 0.0132
Statistical Analysis 10: Comparison: QMF149 150/320 μg vs MF 800 μg; Day 1: 1 hour; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.178, 95% CI 2-sided [0.150 to 0.205], Standard Error of Mean 0.0139
Statistical Analysis 11: Comparison: QMF149 150/160 μg vs MF 400 μg; Day 1: 1hour; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.205, 95% CI 2-sided [0.177 to 0.232], Standard Error of Mean 0.0139
Statistical Analysis 12: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Day 1: 1hour; Test type: Superiority; p = 0.632, MMRM; LS Mean = 0.007, 95% CI 2-sided [-0.021 to 0.034], Standard Error of Mean 0.0139
Statistical Analysis 13: Comparison: QMF149 150/320 μg vs MF 800 μg; Day 30: 5 minutes; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.189, 95% CI 2-sided [0.151 to 0.226], Standard Error of Mean 0.0192
Statistical Analysis 14: Comparison: QMF149 150/160 μg vs MF 400 μg; Day 30: 5 minutes; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.232, 95% CI 2-sided [0.194 to 0.270], Standard Error of Mean 0.0194
Statistical Analysis 15: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Day 30: 5 minutes; Test type: Superiority; p = 0.005, MMRM; LS Mean = 0.053, 95% CI 2-sided [0.016 to 0.091], Standard Error of Mean 0.0191
Statistical Analysis 16: Comparison: QMF149 150/320 μg vs MF 800 μg; Day 30: 30 minutes; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.194, 95% CI 2-sided [0.156 to 0.232], Standard Error of Mean 0.0194
Statistical Analysis 17: Comparison: QMF149 150/160 μg vs MF 400 μg; Day 30: 30 minutes; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.253, 95% CI 2-sided [0.214 to 0.291], Standard Error of Mean 0.0196
Statistical Analysis 18: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Day 30: 30 minutes; Test type: Superiority; p = 0.026, MMRM; LS Mean = 0.043, 95% CI 2-sided [0.005 to 0.08], Standard Error of Mean 0.0192
Statistical Analysis 19: Comparison: QMF149 150/320 μg vs MF 800 μg; Day 30: 1 hour; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.190, 95% CI 2-sided [0.152 to 0.229], Standard Error of Mean 0.0196
Statistical Analysis 20: Comparison: QMF149 150/160 μg vs MF 400 μg; Day 30: 1 hour; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.258, 95% CI 2-sided [0.219 to 0.296], Standard Error of Mean 0.0198
Statistical Analysis 21: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Day 30: 1 hour; Test type: Superiority; p = 0.059, MMRM; LS Mean = 0.037, 95% CI 2-sided [-0.001 to 0.075], Standard Error of Mean 0.0194
Statistical Analysis 22: Comparison: QMF149 150/320 μg vs MF 800 μg; Day 86: 5 minutes; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.163, 95% CI 2-sided [0.123 to 0.203], Standard Error of Mean 0.0204
Statistical Analysis 23: Comparison: QMF149 150/160 μg vs MF 400 μg; Day 86: 5 minutes; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.231, 95% CI 2-sided [0.191 to 0.271], Standard Error of Mean 0.0206
Statistical Analysis 24: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Day 86: 5minutes; Test type: Superiority; p = 0.007, MMRM; LS Mean = 0.055, 95% CI 2-sided [0.015 to 0.095], Standard Error of Mean 0.0203
Statistical Analysis 25: Comparison: QMF149 150/320 μg vs MF 800 μg; Day 86: 30 minutes; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.180, 95% CI 2-sided [0.140 to 0.219], Standard Error of Mean 0.0203
Statistical Analysis 26: Comparison: QMF149 150/160 μg vs MF 400 μg; Day 86: 30 minutes; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.252, 95% CI 2-sided [0.211 to 0.292], Standard Error of Mean 0.0205
Statistical Analysis 27: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Day 86: 30 minutes; Test type: Superiority; p = 0.057, MMRM; LS Mean = 0.038, 95% CI 2-sided [-0.001 to 0.078], Standard Error of Mean 0.0202
Statistical Analysis 28: Comparison: QMF149 150/320 μg vs MF 800 μg; Day 86: 1 hour; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.187, 95% CI 2-sided [0.147 to 0.227], Standard Error of Mean 0.0205
Statistical Analysis 29: Comparison: QMF149 150/160 μg vs MF 400 μg; Day 86: 1 hour; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.249, 95% CI 2-sided [0.208 to 0.289], Standard Error of Mean 0.0208
Statistical Analysis 30: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Day 86: 1hour; Test type: Superiority; p = 0.037, MMRM; LS Mean = 0.043, 95% CI 2-sided [0.003 to 0.083], Standard Error of Mean 0.0205
Statistical Analysis 31: Comparison: QMF149 150/320 μg vs MF 800 μg; Day 183: 5 minutes; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.163, 95% CI 2-sided [0.121 to 0.206], Standard Error of Mean 0.0217
Statistical Analysis 32: Comparison: QMF149 150/160 μg vs MF 400 μg; Day 183: 5 minutes; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.243, 95% CI 2-sided [0.200 to 0.286], Standard Error of Mean 0.0219
Statistical Analysis 33: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Day 183: 5 minutes; Test type: Superiority; p = 0.041, MMRM; LS Mean = 0.044, 95% CI 2-sided [0.002 to 0.087], Standard Error of Mean 0.0216
Statistical Analysis 34: Comparison: QMF149 150/320 μg vs MF 800 μg; Day 183: 30 minutes; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.176, 95% CI 2-sided [0.133 to 0.220], Standard Error of Mean 0.0222
Statistical Analysis 35: Comparison: QMF149 150/160 μg vs MF 400 μg; Day 183: 30 minutes; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.259, 95% CI 2-sided [0.215 to 0.303], Standard Error of Mean 0.0224
Statistical Analysis 36: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Day 183: 30 minutes; Test type: Superiority; p = 0.071, MMRM; LS Mean = 0.04, 95% CI 2-sided [-0.003 to 0.083], Standard Error of Mean 0.0221
Statistical Analysis 37: Comparison: QMF149 150/320 μg vs MF 800 μg; Day 183: 1 hour; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.180, 95% CI 2-sided [0.137 to 0.223], Standard Error of Mean 0.0219
Statistical Analysis 38: Comparison: QMF149 150/160 μg vs MF 400 μg; Day 183: 1 hour; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.259, 95% CI 2-sided [0.215 to 0.302], Standard Error of Mean 0.0222
Statistical Analysis 39: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Day 183: 1 hour; Test type: Superiority; p = 0.071, MMRM; LS Mean = 0.039, 95% CI 2-sided [-0.003 to 0.082], Standard Error of Mean 0.0218
Statistical Analysis 40: Comparison: QMF149 150/320 μg vs MF 800 μg; Day 364: 5 minutes; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.139, 95% CI 2-sided [0.094 to 0.184], Standard Error of Mean 0.0229
Statistical Analysis 41: Comparison: QMF149 150/160 μg vs MF 400 μg; Day 364: 5 minutes; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.249, 95% CI 2-sided [0.205 to 0.294], Standard Error of Mean 0.0228
Statistical Analysis 42: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Day 364: 5 minutes; Test type: Superiority; p = 0.244, MMRM; LS Mean = 0.026, 95% CI 2-sided [-0.018 to 0.071], Standard Error of Mean 0.0227
Statistical Analysis 43: Comparison: QMF149 150/320 μg vs MF 800 μg; Day 364: 30 minutes; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.155, 95% CI 2-sided [0.110 to 0.200], Standard Error of Mean 0.0228
Statistical Analysis 44: Comparison: QMF149 150/160 μg vs MF 400 μg; Day 364: 30 minutes; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.264, 95% CI 2-sided [0.219 to 0.308], Standard Error of Mean 0.0227
Statistical Analysis 45: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Day 364: 30 minutes; Test type: Superiority; p = 0.162, MMRM; LS Mean = 0.032, 95% CI 2-sided [-0.013 to 0.076], Standard Error of Mean 0.0226
Statistical Analysis 46: Comparison: QMF149 150/320 μg vs MF 800 μg; Day 364: 1 hour; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.163, 95% CI 2-sided [0.117 to 0.209], Standard Error of Mean 0.0234
Statistical Analysis 47: Comparison: QMF149 150/160 μg vs MF 400 μg; Day 364: 1 hour; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.262, 95% CI 2-sided [0.216 to 0.308], Standard Error of Mean 0.0232
Statistical Analysis 48: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Day 364: 1 hour; Test type: Superiority; p = 0.182, MMRM; LS Mean = 0.031, 95% CI 2-sided [-0.014 to 0.076], Standard Error of Mean 0.0231

6. Secondary Outcome: Trough Forced Vital Capacity (FVC)
Description: FVC is the total amount of air exhaled during the FEV test. Trough FVC is defined as average of the two FVC measurements taken 23 hr 15 min and 23 hr 45 min post-evening dose. It was assessed by performing spirometric assessment.
Time Frame: Up to Week 52 (Day 365)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | QMF149 150/320 μg | QMF149 150/160 μg | MF 800 μg | MF 400 μg | Salmeterol/Fluticasone 50/500 μg
Number analyzed (Participants) | 439 | 433 | 436 | 441 | 441
L
  Day 2: number analyzed (Participants) | 432 | 430 | 410 | 435 | 419
  Day 2 | 3.342 (0.0173) | 3.342 (0.0174) | 3.256 (0.0177) | 3.203 (0.0173) | 3.344 (0.0176)
  Day 184: number analyzed (Participants) | 395 | 389 | 372 | 376 | 391
  Day 184 | 3.372 (0.0179) | 3.387 (0.0180) | 3.322 (0.0183) | 3.246 (0.0182) | 3.355 (0.0180)
  Day 365: number analyzed (Participants) | 372 | 383 | 365 | 369 | 382
  Day 365 | 3.394 (0.0182) | 3.364 (0.0181) | 3.319 (0.0184) | 3.218 (0.0183) | 3.358 (0.0182)
Statistical Analysis 1: Comparison: QMF149 150/320 μg vs MF 800 μg; Day 2; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.086, 95% CI 2-sided [0.040 to 0.133], Standard Error of Mean 0.0237
Statistical Analysis 2: Comparison: QMF149 150/160 μg vs MF 400 μg; Day 2; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.139, 95% CI 2-sided [0.093 to 0.185], Standard Error of Mean 0.0235
Statistical Analysis 3: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Day 2; Test type: Superiority; p = 0.927, MMRM; LS Mean = -0.002, 95% CI 2-sided [-0.049 to 0.044], Standard Error of Mean 0.0237
Statistical Analysis 4: Comparison: QMF149 150/320 μg vs MF 800 μg; Day 184; Test type: Superiority; p = 0.044, MMRM; LS Mean = 0.050, 95% CI 2-sided [0.001 to 0.098], Standard Error of Mean 0.0246
Statistical Analysis 5: Comparison: QMF149 150/160 μg vs MF 400 μg; Day 184; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.141, 95% CI 2-sided [0.093 to 0.190], Standard Error of Mean 0.0246
Statistical Analysis 6: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Day 184; Test type: Superiority; p = 0.490, MMRM; LS Mean = 0.017, 95% CI 2-sided [-0.031 to 0.065], Standard Error of Mean 0.0244
Statistical Analysis 7: Comparison: QMF149 150/320 μg vs MF 800 μg; Day 365; Test type: Superiority; p = 0.002, MMRM; LS Mean = 0.076, 95% CI 2-sided [0.027 to 0.125], Standard Error of Mean 0.0249
Statistical Analysis 8: Comparison: QMF149 150/160 μg vs MF 400 μg; Day 365; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.146, 95% CI 2-sided [0.098 to 0.195], Standard Error of Mean 0.0248
Statistical Analysis 9: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Day 365; Test type: Superiority; p = 0.143, MMRM; LS Mean = 0.036, 95% CI 2-sided [-0.012 to 0.085], Standard Error of Mean 0.0248

7. Secondary Outcome: Trough Forced Expiratory Flow (FEF)Between 25% and 75% of FVC (FEF25-75)
Description: FEF is the flow (or speed) of air coming out of the lung during the middle portion of a forced expiration. Trough FEF25-75% is defined as average of the two FEF25-75% measurements taken 23 hr 15 min and 23 hr 45 min post-evening dose. It was assessed by performing spirometric assessment.
Time Frame: Up to Week 52 (Day 365)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Litres/second (L/s)
Arm/Group | QMF149 150/320 μg | QMF149 150/160 μg | MF 800 μg | MF 400 μg | Salmeterol/Fluticasone 50/500 μg
Number analyzed (Participants) | 439 | 433 | 436 | 441 | 441
Litres/second (L/s)
  Day 2: number analyzed (Participants) | 432 | 430 | 410 | 435 | 419
  Day 2 | 1.644 (0.0186) | 1.617 (0.0187) | 1.455 (0.0191) | 1.406 (0.0186) | 1.662 (0.0189)
  Day 184: number analyzed (Participants) | 395 | 389 | 372 | 376 | 391
  Day 184 | 1.775 (0.0249) | 1.738 (0.0250) | 1.546 (0.0253) | 1.473 (0.0254) | 1.692 (0.0250)
  Day 365: number analyzed (Participants) | 372 | 383 | 365 | 369 | 382
  Day 365 | 1.745 (0.0259) | 1.686 (0.0257) | 1.530 (0.0261) | 1.440 (0.0261) | 1.692 (0.0258)
Statistical Analysis 1: Comparison: QMF149 150/320 μg vs MF 800 μg; Day 2; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.189, 95% CI 2-sided [0.139 to 0.238], Standard Error of Mean 0.0253
Statistical Analysis 2: Comparison: QMF149 150/160 μg vs MF 400 μg; Day 2; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.210, 95% CI 2-sided [0.161 to 0.259], Standard Error of Mean 0.025
Statistical Analysis 3: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Day 2; Test type: Superiority; p = 0.475, MMRM; LS Mean = -0.018, 95% CI 2-sided [-0.067 to 0.031], Standard Error of Mean 0.0252
Statistical Analysis 4: Comparison: QMF149 150/320 μg vs MF 800 μg; Day 184; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.228, 95% CI 2-sided [0.161 to 0.296], Standard Error of Mean 0.0345
Statistical Analysis 5: Comparison: QMF149 150/160 μg vs MF 400 μg; Day 184; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.265, 95% CI 2-sided [0.197 to 0.333], Standard Error of Mean 0.0346
Statistical Analysis 6: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Day 184; Test type: Superiority; p = 0.015, MMRM; LS Mean = 0.083, 95% CI 2-sided [0.016 to 0.151], Standard Error of Mean 0.0343
Statistical Analysis 7: Comparison: QMF149 150/320 μg vs MF 800 μg; Day 365; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.215, 95% CI 2-sided [0.145 to 0.285], Standard Error of Mean 0.0358
Statistical Analysis 8: Comparison: QMF149 150/160 μg vs MF 400 μg; Day 365; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.246, 95% CI 2-sided [0.176 to 0.316], Standard Error of Mean 0.0357
Statistical Analysis 9: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Day 365; Test type: Superiority; p = 0.139, MMRM; LS Mean = 0.053, 95% CI 2-sided [-0.017 to 0.122], Standard Error of Mean 0.0356

8. Secondary Outcome: Change From Baseline in Morning and Evening Peak Expiratory Flow Rate (PEF) Over 26 and 52 Weeks of Treatment
Description: PEF is a person's maximum speed of expiration. All the participants were instructed to record PEF twice daily using a mini Peak Flow Meter device, once in the morning (before taking the morning dose) and once approximately 12 h later in the evening (before taking the evening dose). At each timepoint, the participant was instructed to perform 3 consecutive manoeuvres within 10 minutes. These PEF values were captured in the e-PEF/diary. The best of 3 values were used.
Time Frame: Up to Weeks 26 and 52
Population: Full Analysis Set (FAS) consisted of all patients in the RAN set who received at least one dose of study medication. n represents tthe number of participants with data at respective visit.
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | QMF149 150/320 μg | QMF149 150/160 μg | MF 800 μg | MF 400 μg | Salmeterol/Fluticasone 50/500 μg
Number analyzed (Participants) | 443 | 437 | 440 | 443 | 444
L/min
  Week 26: Mean morning PEF: number analyzed (Participants) | 418 | 419 | 430 | 422 | 426
  Week 26: Mean morning PEF | 42.4 (2.15) | 38.1 (2.15) | 12.8 (2.13) | 5.9 (2.14) | 29.1 (2.14)
  Week 26:Mean evening PEF: number analyzed (Participants) | 417 | 420 | 425 | 419 | 423
  Week 26:Mean evening PEF | 32.5 (2.05) | 30.4 (2.04) | 7.7 (2.04) | 0.0 (2.05) | 23.9 (2.04)
  Week 52:Mean morning PEF: number analyzed (Participants) | 415 | 420 | 427 | 422 | 424
  Week 52:Mean morning PEF | 42.1 (2.24) | 36.9 (2.22) | 13.4 (2.21) | 6.7 (2.22) | 28.3 (2.22)
  Week 52:Mean evening PEF: number analyzed (Participants) | 416 | 420 | 424 | 418 | 422
  Week 52:Mean evening PEF | 31.2 (2.14) | 28.7 (2.13) | 7.4 (2.13) | -0.3 (2.14) | 22.1 (2.13)
Statistical Analysis 1: Comparison: QMF149 150/320 μg vs MF 800 μg; Week 26: Mean morning PEF; Test type: Superiority; p < 0.001, Linear Mixed Model (LMM); LS Mean = 29.6, 95% CI 2-sided [23.8 to 35.4], Standard Error of Mean 2.96
Statistical Analysis 2: Comparison: QMF149 150/160 μg vs MF 400 μg; Week 26: Mean morning PEF; Test type: Superiority; p < 0.001, LMM; LS Mean = 32.2, 95% CI 2-sided [26.4 to 38.1], Standard Error of Mean 2.97
Statistical Analysis 3: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Week 26: Mean morning PEF; Test type: Superiority; p < 0.001, LMM; LS Mean = 13.3, 95% CI 2-sided [7.5 to 19.1], Standard Error of Mean 2.97
Statistical Analysis 4: Comparison: QMF149 150/320 μg vs MF 800 μg; Week 26: Mean evening PEF; Test type: Superiority; p < 0.001, LMM; LS Mean = 24.8, 95% CI 2-sided [19.3 to 30.3], Standard Error of Mean 2.82
Statistical Analysis 5: Comparison: QMF149 150/160 μg vs MF 400 μg; Week 26: Mean evening PEF; Test type: Superiority; p < 0.001, LMM; LS Mean = 30.4, 95% CI 2-sided [24.8 to 35.9], Standard Error of Mean 2.83
Statistical Analysis 6: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Week 26: Mean evening PEF; Test type: Superiority; p = 0.002, LMM; LS Mean = 8.6, 95% CI 2-sided [3.1 to 14.2], Standard Error of Mean 2.83
Statistical Analysis 7: Comparison: QMF149 150/320 μg vs MF 800 μg; Week 52: Mean morning PEF; Test type: Superiority; p < 0.001, LMM; LS Mean = 28.7, 95% CI 2-sided [22.7 to 34.8], Standard Error of Mean 3.07
Statistical Analysis 8: Comparison: QMF149 150/160 μg vs MF 400 μg; Week 52: Mean morning PEF; Test type: Superiority; p < 0.001, LMM; LS Mean = 30.2, 95% CI 2-sided [24.2 to 36.3], Standard Error of Mean 3.07
Statistical Analysis 9: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Week 52: Mean morning PEF; Test type: Superiority; p < 0.001, LMM; LS Mean = 13.8, 95% CI 2-sided [7.7 to 19.8], Standard Error of Mean 3.08
Statistical Analysis 10: Comparison: QMF149 150/320 μg vs MF 800 μg; Week 52: Mean evening PEF; Test type: Superiority; p < 0.001, LMM; LS Mean = 23.7, 95% CI 2-sided [18.0 to 29.5], Standard Error of Mean 2.94
Statistical Analysis 11: Comparison: QMF149 150/160 μg vs MF 400 μg; Week 52: Mean evening PEF; Test type: Superiority; p < 0.001, LMM; LS Mean = 29.1, 95% CI 2-sided [23.3 to 34.8], Standard Error of Mean 2.94
Statistical Analysis 12: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Week 52: Mean evening PEF; Test type: Superiority; p = 0.002, LMM; LS Mean = 9.1, 95% CI 2-sided [3.3 to 14.9], Standard Error of Mean 2.95

9. Secondary Outcome: Percentage of Participants Achieving the Minimal Important Difference (MID) ACQ ≥ 0.5 at Weeks 26 and 52
Description: Change from baseline in ACQ-7 scores of ≤ 0.5 was defined as minimal clinically important difference and were considered clinically meaningful. The ACQ-7 measured asthma symptom control and consists of 7 items: 5 on symptom assessment, 1 on rescue bronchodilator use and 1 on airway calibre (FEV1 % predicted). All 7 questions of the ACQ-7 were equally weighted. Items 1-5 were scored along a 7-point response scale, where 0 = totally controlled and 6 = severely uncontrolled. Item 6 is scored between 0 = no rescue medication and 6 = More than 16 puffs/inhalations most days. The 7th item was scored by the investigator based on the FEV1 % predicted from the masterscope at the site (i.e., Score = 0 means > 95% of predicted FEV1, 1 = 90 - 95%, 2 = 80 - 89%, 3 = 70 - 79%, 4 = 60 - 69%, 5 = 50 - 59%, and Score = 6 means < 50% of predicted FEV1). The total score was calculated as the mean of all questions
Time Frame: Weeks 26 (Day 183) and 52 (Day 364)
Population: FAS consisted of all participants in the RAN set who received at least one dose of study medication. n represents number of participants with data at the respective visit.
Measure: Number; unit: percentage of participants
Arm/Group | QMF149 150/320 μg | QMF149 150/160 μg | MF 800 μg | MF 400 μg | Salmeterol/Fluticasone 50/500 μg
Number analyzed (Participants) | 442 | 437 | 440 | 443 | 444
percentage of participants
  Day 183: number analyzed (Participants) | 407 | 407 | 405 | 393 | 410
  Day 183 | 76.4 | 76.2 | 72.3 | 66.9 | 75.9
  Day 364: number analyzed (Participants) | 385 | 397 | 387 | 377 | 405
  Day 364 | 77.7 | 82.1 | 73.6 | 69.2 | 77.3
Statistical Analysis 1: Comparison: QMF149 150/320 μg vs QMF149 150/160 μg vs MF 800 μg; Day 183; Test type: Superiority; p = 0.094, Logistic regression model; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.95 to 1.81]
Statistical Analysis 2: Comparison: QMF149 150/160 μg vs MF 400 μg; Day 183; Test type: Superiority; p < 0.001, Logistic regression model; Odds Ratio (OR) = 1.73, 95% CI 2-sided [1.26 to 2.37]
Statistical Analysis 3: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Day 183; Test type: Superiority; p = 0.746, Logistic regression model; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.76 to 1.46]
Statistical Analysis 4: Comparison: QMF149 150/320 μg vs MF 800 μg; Day 364; Test type: Superiority; p = 0.088, Logistic regression model; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.96 to 1.87]
Statistical Analysis 5: Comparison: QMF149 150/160 μg vs MF 400 μg; Day 364; Test type: Superiority; p < 0.001, Logistic regression model; Odds Ratio (OR) = 2.24, 95% CI 2-sided [1.58 to 3.17]
Statistical Analysis 6: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Day 364; Test type: Superiority; p = 0.771, Logistic regression model; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.75 to 1.49]

10. Secondary Outcome: Change From Baseline in Percentage of Asthma Symptoms Free Days
Description: All participants were provided with an electronic diary (e-Diary) to record clinical symptoms. They were instructed to routinely complete the e-Diary twice daily at the same time each morning and again approximately 12 hours later in the evening. The e-Diary was reviewed at each visit until study completion. Asthma symptoms free days are days with no daytime symptoms, no night-time awakenings and no symptoms on awakening. The daytime asthma symptom score was based on the daily e-diary recordings by participants with respect to shortness of breath, wheeze, cough, chest tightness, and impact on usual daily activities due to symptoms.
Time Frame: Up to Week 52
Population: FAS consisted of all participants in the RAN set who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | QMF149 150/320 μg | QMF149 150/160 μg | MF 800 μg | MF 400 μg | Salmeterol/Fluticasone 50/500 μg
Number analyzed (Participants) | 401 | 402 | 408 | 404 | 405
percentage of days | 28.3 (1.72) | 28.4 (1.72) | 22.5 (1.72) | 19.3 (1.72) | 24.9 (1.72)
Statistical Analysis 1: Comparison: QMF149 150/320 μg vs MF 800 μg; Test type: Superiority; p = 0.012, Linear Mixed Model (LMM); LS Mean = 5.8, 95% CI 2-sided [1.3 to 10.2], Standard Error of Mean 2.29
Statistical Analysis 2: Comparison: QMF149 150/160 μg vs MF 400 μg; Test type: Superiority; p < 0.001, LMM; LS Mean = 9.1, 95% CI 2-sided [4.6 to 13.6], Standard Error of Mean 2.29
Statistical Analysis 3: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Test type: Superiority; p = 0.135, LMM; LS Mean = 3.4, 95% CI 2-sided [-1.1 to 7.9], Standard Error of Mean 2.29

11. Secondary Outcome: Change Form Baseline in Percentage of Days With no Daytime Symptoms
Description: All participants were provided with an electronic diary (e-Diary) to record clinical symptoms. They were instructed to routinely complete the e-Diary twice daily at the same time each morning and again approximately 12 hours later in the evening. The e-Diary was reviewed at each visit until study completion. For days with no daytime symptoms, all 5 evening questions must have a score = 0 with respect to shortness of breath, wheeze, cough, chest tightness and impact on usual daily activities due to symptoms, each with scores from 0 (no problems) to 4 (very severe problems).
Time Frame: Up to Week 52
Population: FAS consisted of all participants in the RAN set who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | QMF149 150/320 μg | QMF149 150/160 μg | MF 800 μg | MF 400 μg | Salmeterol/Fluticasone 50/500 μg
Number analyzed (Participants) | 416 | 420 | 425 | 419 | 423
percentage of days | 28.0 (1.69) | 28.0 (1.69) | 23.0 (1.68) | 20.0 (1.69) | 24.8 (1.68)
Statistical Analysis 1: Comparison: QMF149 150/320 μg vs MF 800 μg; Test type: Superiority; p = 0.026, LMM; LS Mean = 5.0, 95% CI 2-sided [0.6 to 9.4], Standard Error of Mean 2.25
Statistical Analysis 2: Comparison: QMF149 150/160 μg vs MF 400 μg; Test type: Superiority; p < 0.001, LMM; LS Mean = 8.1, 95% CI 2-sided [3.7 to 12.5], Standard Error of Mean 2.25
Statistical Analysis 3: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Test type: Superiority; p = 0.151, LMM; LS Mean = 3.2, 95% CI 2-sided [-1.2 to 7.7], Standard Error of Mean 2.25

12. Secondary Outcome: Change From Baseline in Percentage of Nights With no Night-time Awakenings
Description: All participants were provided with an electronic diary (e-Diary) to record clinical symptoms. They were instructed to routinely complete the e-Diary twice daily at the same time each morning and again approximately 12 hours later in the evening. The e-Diary was reviewed at each visit until study completion. The question asked for nights with no night-time awakenings was "How did you sleep last night?" had to be answered with "I did not wake up because of any breathing problems" with scores from 0 (no problem)-4 (very severe problems).
Time Frame: Up to Week 52
Population: FAS consisted of all participants in the RAN set who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: percentage of nights
Arm/Group | QMF149 150/320 μg | QMF149 150/160 μg | MF 800 μg | MF 400 μg | Salmeterol/Fluticasone 50/500 μg
Number analyzed (Participants) | 415 | 420 | 428 | 422 | 424
percentage of nights | 17.0 (1.28) | 16.4 (1.27) | 14.2 (1.27) | 12.5 (1.27) | 16.1 (1.27)
Statistical Analysis 1: Comparison: QMF149 150/320 μg vs MF 800 μg; Test type: Superiority; p = 0.104, LMM; LS Mean = 2.8, 95% CI 2-sided [-0.6 to 6.2], Standard Error of Mean 1.72
Statistical Analysis 2: Comparison: QMF149 150/160 μg vs MF 400 μg; Test type: Superiority; p = 0.024, LMM; LS Mean = 3.9, 95% CI 2-sided [0.5 to 7.3], Standard Error of Mean 1.72
Statistical Analysis 3: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Test type: Superiority; p = 0.588, LMM; LS Mean = 0.9, 95% CI 2-sided [-2.5 to 4.3], Standard Error of Mean 1.73

13. Secondary Outcome: Change Form Baseline in Percentage of Mornings With no Symptoms on Awakening
Description: All participants were provided with an electronic diary (e-Diary) to record clinical symptoms. They were instructed to routinely complete the e-Diary twice daily at the same time each morning and again approximately 12 hours later in the evening. The e-Diary was reviewed at each visit until study completion. The question asked for mornings with no symptoms on awakening was "Did you have asthma symptoms upon awakening in the morning?" to be answered with "None" with scores from 0 (no problem)-4 (very severe problems).
Time Frame: Up to Week 52
Population: FAS consisted of all participants in the RAN set who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: percentage of mornings
Arm/Group | QMF149 150/320 μg | QMF149 150/160 μg | MF 800 μg | MF 400 μg | Salmeterol/Fluticasone 50/500 μg
Number analyzed (Participants) | 415 | 420 | 428 | 422 | 424
percentage of mornings | 25.5 (1.66) | 22.9 (1.65) | 19.1 (1.65) | 14.1 (1.65) | 20.7 (1.65)
Statistical Analysis 1: Comparison: QMF149 150/320 μg vs MF 800 μg; Test type: Superiority; p = 0.003, LMM; LS Mean = 6.4, 95% CI 2-sided [2.1 to 10.7], Standard Error of Mean 2.19
Statistical Analysis 2: Comparison: QMF149 150/160 μg vs MF 400 μg; Test type: Superiority; p < 0.001, LMM; LS Mean = 8.9, 95% CI 2-sided [4.6 to 13.2], Standard Error of Mean 2.19
Statistical Analysis 3: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Test type: Superiority; p = 0.029, LMM; LS Mean = 4.8, 95% CI 2-sided [0.5 to 9.1], Standard Error of Mean 2.2

14. Secondary Outcome: Rescue Medication Usage
Description: All participants were given salbutamol/albuterol to use as rescue medication throughout the study along with e-Diary to record rescue medication use. The number of puffs of rescue medication during the past 12 hours is recorded twice (morning/evening) by the participant prior to taking study medication. The mean daily number of puffs of rescue medication use will be calculated for each participant, done separately for morning (night-time), evening (daytime), and daily (night-time plus daytime) rescue medication use
Time Frame: Up to Weeks 26 and 52
Population: FAS consisted of all participants in the RAN set who received at least one dose of study medication. n represents number of participants included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: number of puffs
Arm/Group | QMF149 150/320 μg | QMF149 150/160 μg | MF 800 μg | MF 400 μg | Salmeterol/Fluticasone 50/500 μg
Number analyzed (Participants) | 443 | 437 | 440 | 443 | 444
number of puffs
  Week1-26 Mean night-time number of puffs: number analyzed (Participants) | 418 | 419 | 430 | 422 | 426
  Week1-26 Mean night-time number of puffs | -0.38 (0.028) | -0.27 (0.028) | -0.26 (0.028) | -0.19 (0.028) | -0.34 (0.028)
  Week1-26 Mean daytime number of puffs: number analyzed (Participants) | 417 | 420 | 427 | 419 | 424
  Week1-26 Mean daytime number of puffs | -0.57 (0.035) | -0.46 (0.035) | -0.38 (0.035) | -0.34 (0.035) | -0.53 (0.035)
  Week1-26 Mean daily number of puffs: number analyzed (Participants) | 426 | 428 | 433 | 428 | 432
  Week1-26 Mean daily number of puffs | -0.96 (0.059) | -0.73 (0.059) | -0.65 (0.059) | -0.53 (0.059) | -0.87 (0.059)
  Week1-52 Mean night-time number of puffs: number analyzed (Participants) | 415 | 420 | 428 | 422 | 424
  Week1-52 Mean night-time number of puffs | -0.40 (0.029) | -0.30 (0.029) | -0.29 (0.028) | -0.20 (0.029) | -0.35 (0.029)
  Week 1-52 Mean daytime number of puffs: number analyzed (Participants) | 416 | 420 | 425 | 419 | 423
  Week 1-52 Mean daytime number of puffs | -0.60 (0.035) | -0.51 (0.035) | -0.43 (0.035) | -0.36 (0.035) | -0.55 (0.035)
  Week 1-52 Mean daily number of puffs: number analyzed (Participants) | 426 | 428 | 433 | 428 | 432
  Week 1-52 Mean daily number of puffs | -1.00 (0.060) | -0.80 (0.060) | -0.72 (0.060) | -0.56 (0.060) | -0.91 (0.060)
Statistical Analysis 1: Comparison: QMF149 150/320 μg vs MF 800 μg; Week1-26 Mean night-time number of puffs; Test type: Superiority; p = 0.001, LMM; LS Mean = -0.13, 95% CI 2-sided [-0.2 to -0.05], Standard Error of Mean 0.039
Statistical Analysis 2: Comparison: QMF149 150/160 μg vs MF 400 μg; Week 1-26 Mean night-time number of puffs; Test type: Superiority; p = 0.035, LMM; LS Mean = -0.08, 95% CI 2-sided [-0.16 to -0.01], Standard Error of Mean 0.039
Statistical Analysis 3: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Week 1-26 Mean night-time number of puffs; Test type: Superiority; p = 0.261, LMM; LS Mean = -0.04, 95% CI 2-sided [-0.12 to 0.03], Standard Error of Mean 0.039
Statistical Analysis 4: Comparison: QMF149 150/320 μg vs MF 800 μg; Week 1-26 Mean daytime number of puffs; Test type: Superiority; p < 0.001, LMM; LS Mean = -0.19, 95% CI 2-sided [-0.28 to -0.09], Standard Error of Mean 0.047
Statistical Analysis 5: Comparison: QMF149 150/160 μg vs MF 400 μg; Week 1-26 Mean daytime number of puffs; Test type: Superiority; p = 0.011, LMM; LS Mean = -0.12, 95% CI 2-sided [-0.21 to -0.03], Standard Error of Mean 0.047
Statistical Analysis 6: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Week 1-26 Mean daytime number of puffs; Test type: Superiority; p = 0.425, LMM; LS Mean = -0.04, 95% CI 2-sided [-0.13 to 0.06], Standard Deviation 0.047
Statistical Analysis 7: Comparison: QMF149 150/320 μg vs MF 800 μg; Week 1-26 Mean daily number of puffs; Test type: Superiority; p < 0.001, LMM; LS Mean = -0.31, 95% CI 2-sided [-0.46 to -0.15], Standard Error of Mean 0.081
Statistical Analysis 8: Comparison: QMF149 150/160 μg vs MF 400 μg; Week 1-26 Mean daily number of puffs; Test type: Superiority; p = 0.017, LMM; LS Mean = -0.19, 95% CI 2-sided [-0.35 to -0.03], Standard Error of Mean 0.081
Statistical Analysis 9: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Week 1-26 Mean daily number of puffs; Test type: Superiority; p = 0.29, LMM; LS Mean = -0.09, 95% CI 2-sided [-0.24 to -0.07], Standard Error of Mean 0.081
Statistical Analysis 10: Comparison: QMF149 150/320 μg vs MF 800 μg; Week 1-52 Mean night-time number of puffs; Test type: Superiority; p = 0.004, LMM; LS Mean = -0.11, 95% CI 2-sided [-0.19 to -0.04], Standard Error of Mean 0.039
Statistical Analysis 11: Comparison: QMF149 150/160 μg vs MF 400 μg; Week 1-52 Mean night-time number of puffs; Test type: Superiority; p = 0.019, LMM; LS Mean = -0.09, 95% CI 2-sided [-0.17 to -0.02], Standard Error of Mean 0.039
Statistical Analysis 12: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Week 1-52 Mean night-time number of puffs; Test type: Superiority; p = 0.226, LMM; LS Mean = -0.05, 95% CI 2-sided [-0.12 to 0.03], Standard Error of Mean 0.039
Statistical Analysis 13: Comparison: QMF149 150/320 μg vs MF 800 μg; Week 1-52 Mean daytime number of puffs; Test type: Superiority; p < 0.001, LMM; LS Mean = -0.17, 95% CI 2-sided [-0.26 to -0.07], Standard Error of Mean 0.048
Statistical Analysis 14: Comparison: QMF149 150/160 μg vs MF 400 μg; Week 1-52 Mean daytime number of puffs; Test type: Superiority; p = 0.002, LMM; LS Mean = -0.15, 95% CI 2-sided [-0.24 to -0.05], Standard Error of Mean 0.048
Statistical Analysis 15: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Week 1-52 Mean daytime number of puffs; Test type: Superiority; p = 0.384, LMM; LS Mean = -0.04, 95% CI 2-sided [-0.14 to 0.05], Standard Error of Mean 0.048
Statistical Analysis 16: Comparison: QMF149 150/320 μg vs MF 800 μg; Week 1-52 Mean daily number of puffs; Test type: Superiority; p < 0.001, LMM; LS Mean = -0.28, 95% CI 2-sided [-0.44 to -0.12], Standard Error of Mean 0.081
Statistical Analysis 17: Comparison: QMF149 150/160 μg vs MF 400 μg; Week 1-52 Mean daily number of puffs; Test type: Superiority; p = 0.004, LMM; LS Mean = -0.23, 95% CI 2-sided [-0.39 to -0.07], Standard Error of Mean 0.081
Statistical Analysis 18: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Week 1-52 Mean daily number of puffs; Test type: Superiority; p = 0.245, LMM; LS Mean = -0.09, 95% CI 2-sided [-0.25 to 0.06], Standard Error of Mean 0.081

15. Secondary Outcome: Time to First Asthma Exacerbation by Exacerbation Category
Description: The exacerbation categories were: All (mild, moderate and severe) and combination of moderate or severe and severe.
Time Frame: Up to Week 52
Population: FAS consisted of all participants in the RAN set who received at least one dose of study medication.
Measure: Median (Full Range); unit: days
Arm/Group | QMF149 150/320 μg | QMF149 150/160 μg | MF 800 μg | MF 400 μg | Salmeterol/Fluticasone 50/500 μg
Number analyzed (Participants) | 443 | 437 | 440 | 443 | 444
days
  Moderate or severe asthma exacerbation | 366.0 [2 to 389] | 366.0 [1 to 429] | 366.0 [2 to 390] | 364.0 [2 to 402] | 366.0 [2 to 395]
  Severe asthma exacerbation | 367 [2 to 389] | 366 [1 to 429] | 366 [2 to 390] | 366 [2 to 402] | 366 [3 to 395]
  All (mild, moderate or severe) asthma exacerbation | 366.0 [2 to 389] | 366.0 [1 to 429] | 364.5 [2 to 390] | 306.0 [2 to 402] | 365.0 [2 to 394]
Statistical Analysis 1: Comparison: QMF149 150/320 μg vs MF 800 μg; Moderate or severe asthma exacerbation; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.53, 95% CI 2-sided [0.39 to 0.72]
Statistical Analysis 2: Comparison: QMF149 150/160 μg vs MF 400 μg; Moderate or severe asthma exacerbation; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.45, 95% CI 2-sided [0.34 to 0.6]
Statistical Analysis 3: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Moderate or severe asthma exacerbation; Test type: Superiority; p = 0.209, Regression, Cox; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.59 to 1.12]
Statistical Analysis 4: Comparison: QMF149 150/320 μg vs MF 800 μg; Severe asthma exacerbation; Test type: Superiority; p = 0.003, Regression, Cox; Hazard Ratio (HR) = 0.54, 95% CI 2-sided [0.36 to 0.81]
Statistical Analysis 5: Comparison: QMF149 150/160 μg vs MF 400 μg; Severe asthma exacerbation; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.44, 95% CI 2-sided [0.3 to 0.63]
Statistical Analysis 6: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Severe asthma exacerbation; Test type: Superiority; p = 0.115, Regression, Cox; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.47 to 1.09]
Statistical Analysis 7: Comparison: QMF149 150/320 μg vs MF 800 μg; All asthma exacerbation; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.51 to 0.82]
Statistical Analysis 8: Comparison: QMF149 150/160 μg vs MF 400 μg; All asthma exacerbation; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.48, 95% CI 2-sided [0.38 to 0.6]
Statistical Analysis 9: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; All asthma exacerbation; Test type: Superiority; p = 0.185, Regression, Cox; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.66 to 1.08]

16. Secondary Outcome: Time to First Hospitalization for Asthma Exacerbation
Description: The exacerbation categories were: All (mild, moderate and severe) and combination of moderate or severe and severe.
Time Frame: Up to Week 52
Population: FAS consisted of all participants in the RAN set who received at least one dose of study medication.
Measure: Median (Full Range); unit: days
Arm/Group | QMF149 150/320 μg | QMF149 150/160 μg | MF 800 μg | MF 400 μg | Salmeterol/Fluticasone 50/500 μg
Number analyzed (Participants) | 443 | 437 | 440 | 443 | 444
days | 367.0 [2 to 389] | 367.0 [1 to 429] | 367.0 [2 to 390] | 366.0 [2 to 402] | 367.0 [3 to 395]
Statistical Analysis 1: Comparison: QMF149 150/320 μg vs MF 800 μg; Test type: Superiority; p = 0.337, Regression, Cox; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.13 to 2.03]
Statistical Analysis 2: Comparison: QMF149 150/160 μg vs MF 400 μg; Test type: Superiority; p = 0.063, Regression, Cox; Hazard Ratio (HR) = 0.14, 95% CI 2-sided [0.02 to 1.11]
Statistical Analysis 3: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Test type: Superiority; p = 0.599, Regression, Cox; Hazard Ratio (HR) = 1.62, 95% CI 2-sided [0.27 to 9.7]

17. Secondary Outcome: Annual Rate of Asthma Exacerbations by Exacerbation Category
Description: The exacerbation categories were: All (mild, moderate and severe) and combination of moderate or severe and severe.
Time Frame: Up to Week 52
Population: FAS consisted of all participants in the RAN set who received at least one dose of study medication.
Measure: Mean (95% Confidence Interval); unit: exacerbations per year
Arm/Group | QMF149 150/320 μg | QMF149 150/160 μg | MF 800 μg | MF 400 μg | Salmeterol/Fluticasone 50/500 μg
Number analyzed (Participants) | 443 | 437 | 440 | 443 | 444
exacerbations per year
  Moderate or severe asthma exacerbation | 0.25 [0.20 to 0.32] | 0.27 [0.21 to 0.34] | 0.39 [0.32 to 0.48] | 0.56 [0.46 to 0.68] | 0.27 [0.22 to 0.34]
  Severe asthma exacerbation | 0.13 [0.09 to 0.17] | 0.13 [0.10 to 0.18] | 0.18 [0.13 to 0.23] | 0.29 [0.23 to 0.38] | 0.14 [0.10 to 0.19]
  All (mild, moderate, severe) asthma exacerbation | 0.49 [0.41 to 0.60] | 0.48 [0.40 to 0.59] | 0.74 [0.62 to 0.88] | 1.05 [0.89 to 1.24] | 0.52 [0.43 to 0.63]
Statistical Analysis 1: Comparison: QMF149 150/320 μg vs QMF149 150/160 μg; Moderate or severe asthma exacerbation; Test type: Superiority; p = 0.008, Generalized linear model; Rate Ratio = 0.65, 95% CI 2-sided [0.48 to 0.89]
Statistical Analysis 2: Comparison: QMF149 150/160 μg vs MF 400 μg; Moderate or severe asthma exacerbation; Test type: Superiority; p < 0.001, Generalized linear model; Rate Ratio = 0.47, 95% CI 2-sided [0.35 to 0.64]
Statistical Analysis 3: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Moderate or severe asthma exacerbation; Test type: Superiority; p = 0.669, Generalized linear model; Rate Ratio = 0.93, 95% CI 2-sided [0.67 to 1.29]
Statistical Analysis 4: Comparison: QMF149 150/320 μg vs MF 800 μg; Severe asthma exacerbation; Test type: Superiority; p = 0.108, Generalized linear model; Rate Ratio = 0.71, 95% CI 2-sided [0.47 to 1.08]
Statistical Analysis 5: Comparison: QMF149 150/160 μg vs MF 400 μg; Severe asthma exacerbation; Test type: Superiority; p < 0.001, Generalized linear model; Rate Ratio = 0.46, 95% CI 2-sided [0.31 to 0.67]
Statistical Analysis 6: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Severe asthma exacerbation; Test type: Superiority; p = 0.597, Generalized linear model; Rate Ratio = 0.89, 95% CI 2-sided [0.58 to 1.37]
Statistical Analysis 7: Comparison: QMF149 150/320 μg vs MF 800 μg; All (mild, moderate, severe) asthma exacerbation; Test type: Superiority; p = 0.002, Generalized linear model; Rate Ratio = 0.67, 95% CI 2-sided [0.52 to 0.87]
Statistical Analysis 8: Comparison: QMF149 150/160 μg vs MF 400 μg; All (mild, moderate, severe) asthma exacerbation; Test type: Superiority; p < 0.001, Generalized linear model; Rate Ratio = 0.46, 95% CI 2-sided [0.36 to 0.59]
Statistical Analysis 9: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; All (mild, moderate, severe) asthma exacerbation; Test type: Superiority; p = 0.681, Generalized linear model; Rate Ratio = 0.95, 95% CI 2-sided [0.72 to 1.23]

18. Secondary Outcome: Duration in Days of Asthma Exacerbations by Exacerbation Category
Description: The exacerbation categories were: All (mild, moderate and severe) and combination of moderate or severe and severe.
Time Frame: Up to Week 52
Population: FAS consisted of all participant in the RAN set who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | QMF149 150/320 μg | QMF149 150/160 μg | MF 800 μg | MF 400 μg | Salmeterol/Fluticasone 50/500 μg
Number analyzed (Participants) | 443 | 437 | 440 | 443 | 444
days
  Moderate or severe asthma exacerbation | 2.6 (10.60) | 3.0 (12.53) | 3.7 (11.40) | 5.8 (13.98) | 3.1 (9.68)
  Severe asthma exacerbation | 1.3 (6.02) | 1.7 (8.48) | 1.7 (6.07) | 3.2 (9.16) | 1.9 (7.76)
  All(mild, moderate,severe) asthma exacerbation | 5.4 (18.81) | 5.0 (17.55) | 6.9 (22.96) | 10.1 (25.15) | 5.1 (14.48)
Statistical Analysis 1: Comparison: QMF149 150/320 μg vs MF 800 μg; Moderate or severe asthma exacerbation; Test type: Superiority; p < 0.001, van Elteren test
Statistical Analysis 2: Comparison: QMF149 150/160 μg vs MF 400 μg; Moderate or severe asthma exacerbation; Test type: Superiority; p < 0.001, van Elteren test
Statistical Analysis 3: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Moderate or severe asthma exacerbation; Test type: Superiority; p = 0.059, van Elteren test
Statistical Analysis 4: Comparison: QMF149 150/320 μg vs MF 800 μg; Severe Asthma Exacerbation; Test type: Superiority; p = 0.004, Van Elteren Test
Statistical Analysis 5: Comparison: QMF149 150/160 μg vs MF 400 μg; Severe Asthma Exacerbation; Test type: Superiority; p < 0.001, Van Elteren Test
Statistical Analysis 6: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Severe asthma exacerbation; Test type: Superiority; p = 0.025, van Elteren test
Statistical Analysis 7: Comparison: QMF149 150/320 μg vs MF 800 μg; All(mild, moderate, severe) Asthma Exacerbation; Test type: Superiority; p = 0.002, Van Elteren Test
Statistical Analysis 8: Comparison: QMF149 150/160 μg vs MF 400 μg; All (mild, moderate, severe) Asthma Exacerbation; Test type: Superiority; p < 0.001, Van Elteren Test
Statistical Analysis 9: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; All (mild, moderate, severe) asthma exacerbation; Test type: Superiority; p = 0.074, van Elteren test

19. Secondary Outcome: Percentage of Participants With at Least One Asthma Exacerbation by Exacerbation Category
Description: The exacerbation categories were: All (mild, moderate and severe) and combination of moderate or severe and severe.
Time Frame: Up to Week 52
Population: FAS consisted of all patients in the RAN set who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | QMF149 150/320 μg | QMF149 150/160 μg | MF 800 μg | MF 400 μg | Salmeterol/Fluticasone 50/500 μg
Number analyzed (Participants) | 443 | 437 | 440 | 443 | 444
percentage of participants
  Moderate or severe asthma exacerbation | 14.9 | 16.9 | 26.1 | 32.5 | 19.1
  Severe asthma exacerbation | 8.1 | 9.8 | 14.5 | 20.1 | 11.9
  Moderate asthma exacerbation | 7.7 | 8.2 | 14.3 | 16.5 | 9.2
  Mild asthma exacerbation | 13.3 | 12.1 | 17.5 | 19.6 | 15.1
  All (mild, moderate, severe) asthma exacerbation | 25.5 | 25.6 | 36.1 | 44.5 | 30.6

20. Secondary Outcome: Time in Days to Permanent Discontinuation of Study Medication Due to Asthma Exacerbations
Description: The exacerbation categories were: All (mild, moderate and severe) and combination of moderate or severe and severe.
Time Frame: Up to Week 52
Population: FAS consisted of all participants in the RAN set who received at least one dose of study medication.
Measure: Median (Full Range); unit: days
Arm/Group | QMF149 150/320 μg | QMF149 150/160 μg | MF 800 μg | MF 400 μg | Salmeterol /Fluticasone 50/500 μg
Number analyzed (Participants) | 443 | 437 | 440 | 443 | 444
days | 367.0 [2 to 389] | 367.0 [1 to 429] | 367.0 [2 to 390] | 366.0 [2 to 402] | 367.0 [3 to 395]
Statistical Analysis 1: Comparison: QMF149 150/320 μg vs MF 800 μg; Test type: Superiority; p = 0.222, Regression, Cox; Hazard Ratio (HR) = 0.26, 95% CI 2-sided [0.03 to 2.29]
Statistical Analysis 2: Comparison: QMF149 150/160 μg vs MF 400 μg; Test type: Superiority; p = 0.992, Regression, Cox; Hazard Ratio (HR) = 0, 95% CI 2-sided [lower limit 0] (The upper limit of CI could not be calculated due to low number of participants with asthma exacerbation.)
Statistical Analysis 3: Comparison: QMF149 150/320 μg vs Salmeterol /Fluticasone 50/500 μg; Test type: Superiority; p = 0.618, Regression, Cox; Hazard Ratio (HR) = 0.54, 95% CI 2-sided [0.05 to 6.01]

21. Secondary Outcome: Percentage of Participants Who Permanently Discontinued Study Medication Due to Asthma Exacerbations
Time Frame: Up to Week 52
Population: FAS consisted of all participants in the RAN set who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | QMF149 150/320 μg | QMF149 150/160 μg | MF 800 μg | MF 400 μg | Salmeterol/Fluticasone 50/500 μg
Number analyzed (Participants) | 443 | 437 | 440 | 443 | 444
percentage of participants | 0.2 | 0 | 0.9 | 1.6 | 0.5

22. Secondary Outcome: Total Amounts of Systemic Corticosteroids (in Doses) Used to Treat Asthma Exacerbations
Description: The treatment of asthma exacerbations including the initiation of systemic corticosteroids were done according to investigator's or treating physician's medical judgement and in line with national and international recommendations. If systemic corticosteroids were required, a participant could return to the study after successfully completing a taper of approximately 7-10 days.
Time Frame: Up to Week 52
Population: FAS consisted of all participants in the RAN set who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | QMF149 150/320 μg | QMF149 150/160 μg | MF 800 μg | MF 400 μg | Salmeterol/Fluticasone 50/500 μg
Number analyzed (Participants) | 443 | 437 | 440 | 443 | 444
milligrams | 26.0 (136.92) | 29.9 (124.98) | 28.0 (95.18) | 47.8 (139.98) | 26.9 (114.36)

23. Secondary Outcome: Change From Baseline in Percentage of Rescue Medication Free Days
Description: All participants were given salbutamol/albuterol to use as rescue medication throughout the study along with e-Diary to record rescue medication use. Rescue medication free days is defined as any day where the participant did not use any puffs of rescue medication during daytime and night-time.
Time Frame: Up to Weeks 26 and 52
Population: FAS consisted of all participants in the RAN set who received at least one dose of study medication. n represents number of participants with data at respective visit.
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Groups:
- QMF149 150/320 μg: QMF149 (Indacaterol acetate/Mometasone furoate) 150/320 μg was delivered o.d via Concept1 inhaler in the evening
- QMF149 150/160 μg: QMF149 (Indacaterol acetate/Mometasone furoate) 150/160 μg was delivered o.d via Concept1 inhaler in the evening
Arm/Group | QMF149 150/320 μg | QMF149 150/160 μg | MF 800 μg | MF 400 μg | Salmeterol /Fluticasone 50/500 μg
Number analyzed (Participants) | 443 | 437 | 440 | 443 | 444
percentage of days
  Weeks 1-26: number analyzed (Participants) | 412 | 416 | 424 | 414 | 421
  Weeks 1-26 | 31.5 (1.53) | 27.4 (1.53) | 21.4 (1.52) | 19.1 (1.53) | 27.4 (1.52)
  Weeks 1-52: number analyzed (Participants) | 408 | 416 | 420 | 414 | 416
  Weeks 1-52 | 33.1 (1.55) | 29.4 (1.54) | 23.5 (1.54) | 20.8 (1.54) | 28.8 (1.54)
Statistical Analysis 1: Comparison: QMF149 150/320 μg vs MF 800 μg; Weeks 1-26; Test type: Superiority; p < 0.001, LMM; LS Mean = 10.1, 95% CI 2-sided [6.2 to 14.1], Standard Error of Mean 2.02
Statistical Analysis 2: Comparison: QMF149 150/160 μg vs MF 400 μg; Weeks 1-26; Test type: Superiority; p < 0.001, LMM; LS Mean = 8.3, 95% CI 2-sided [4.3 to 12.3], Standard Error of Mean 2.02
Statistical Analysis 3: Comparison: QMF149 150/320 μg vs Salmeterol /Fluticasone 50/500 μg; Weeks 1-26; Test type: Superiority; p = 0.045, LMM; LS Mean = 4.1, 95% CI 2-sided [0.1 to 8], Standard Error of Mean 2.02
Statistical Analysis 4: Comparison: QMF149 150/320 μg vs MF 800 μg; Weeks 1-52; Test type: Superiority; p < 0.001, LMM; LS Mean = 9.6, 95% CI 2-sided [5.7 to 13.6], Standard Error of Mean 2.03
Statistical Analysis 5: Comparison: QMF149 150/160 μg vs MF 400 μg; Weeks 1-52; Test type: Superiority; p < 0.001, LMM; LS Mean = 8.6, 95% CI 2-sided [4.7 to 12.6], Standard Error of Mean 2.03
Statistical Analysis 6: Comparison: QMF149 150/320 μg vs Salmeterol /Fluticasone 50/500 μg; Weeks 1-52; Test type: Superiority; p = 0.034, LMM; LS Mean = 4.3, 95% CI 2-sided [0.3 to 8.3], Standard Error of Mean 2.04

24. Secondary Outcome: Asthma Quality of Life Questionnaire (AQLQ)
Description: AQLQ is a 32-item disease specific questionnaire designed to measure functional impairments that are most important to patients with asthma, with a recall time of two weeks and each question to be answered on a 7-point scale (1-totally limited/problems all the time, 7-not at all limited/no problems). It consists of 4 domains:
  * Symptoms = Mean of Items 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 29, 30 (12 items)
  * Activity limitation = Mean of Items 1, 2, 3, 4, 5, 11, 19, 25, 28, 31, 32 (11 items)
  * Emotional function = Mean of Items 7, 13, 15, 21, 27 (5 items)
  * Environmental stimuli = Mean of Items 9, 17, 23, 26 (4 items)
  * Overall Score = Mean of Items 1 to 32 (32 items)
Time Frame: Up to Week 52 (Day 364)
Population: FAS consisted of all participants in the RAN set who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | QMF149 150/320 μg | QMF149 150/160 μg | MF 800 μg | MF 400 μg | Salmeterol/Fluticasone 50/500 μg
Number analyzed (Participants) | 428 | 426 | 431 | 428 | 438
score on a scale
  Day 30: number analyzed (Participants) | 427 | 423 | 430 | 425 | 436
  Day 30 | 5.560 (0.0327) | 5.498 (0.0328) | 5.413 (0.0326) | 5.374 (0.0327) | 5.515 (0.0324)
  Day 86: number analyzed (Participants) | 419 | 416 | 422 | 406 | 428
  Day 86 | 5.618 (0.0356) | 5.629 (0.0357) | 5.564 (0.0355) | 5.510 (0.0359) | 5.592 (0.0352)
  Day 183: number analyzed (Participants) | 406 | 407 | 405 | 393 | 410
  Day 183 | 5.724 (0.0372) | 5.738 (0.0372) | 5.598 (0.0372) | 5.581 (0.0376) | 5.639 (0.0369)
  Day 254: number analyzed (Participants) | 392 | 395 | 388 | 385 | 405
  Day 254 | 5.761 (0.0383) | 5.781 (0.0382) | 5.689 (0.0383) | 5.614 (0.0386) | 5.700 (0.0378)
  Day 364: number analyzed (Participants) | 384 | 397 | 389 | 378 | 405
  Day 364 | 5.783 (0.0391) | 5.832 (0.0388) | 5.705 (0.0389) | 5.641 (0.0394) | 5.742 (0.0384)
Statistical Analysis 1: Comparison: QMF149 150/320 μg vs MF 800 μg; Day 30; Test type: Superiority; p = 0.002, MMRM; LS Mean = 0.147, 95% CI 2-sided [0.056 to 0.237], Standard Error of Mean 0.0462
Statistical Analysis 2: Comparison: QMF149 150/160 μg vs MF 400 μg; Day 30; Test type: Superiority; p = 0.008, MMRM; LS Mean = 0.123, 95% CI 2-sided [0.032 to 0.214], Standard Error of Mean 0.0464
Statistical Analysis 3: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Day 30; Test type: Superiority; p = 0.33, MMRM; LS Mean = 0.045, 95% CI 2-sided [-0.045 to 0.135], Standard Error of Mean 0.046
Statistical Analysis 4: Comparison: QMF149 150/320 μg vs MF 800 μg; Day 86; Test type: Superiority; p = 0.28, MMRM; LS Mean = 0.054, 95% CI 2-sided [-0.044 to 0.153], Standard Error of Mean 0.0503
Statistical Analysis 5: Comparison: QMF149 150/160 μg vs MF 400 μg; Day 86; Test type: Superiority; p = 0.02, MMRM; LS Mean = 0.118, 95% CI 2-sided [0.019 to 0.217], Standard Error of Mean 0.0507
Statistical Analysis 6: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Day 86; Test type: Superiority; p = 0.598, MMRM; LS Mean = 0.026, 95% CI 2-sided [-0.072 to 0.125], Standard Error of Mean 0.0501
Statistical Analysis 7: Comparison: QMF149 150/320 μg vs MF 800 μg; Day 183; Test type: Superiority; p = 0.016, MMRM; LS Mean = 0.127, 95% CI 2-sided [0.023 to 0.23], Standard Error of Mean 0.0526
Statistical Analysis 8: Comparison: QMF149 150/160 μg vs MF 400 μg; Day 183; Test type: Superiority; p = 0.003, MMRM; LS Mean = 0.156, 95% CI 2-sided [0.053 to 0.26], Standard Error of Mean 0.0529
Statistical Analysis 9: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Day 183; Test type: Superiority; p = 0.103, MMRM; LS Mean = 0.085, 95% CI 2-sided [-0.017 to 0.188], Standard Error of Mean 0.0525
Statistical Analysis 10: Comparison: QMF149 150/320 μg vs MF 800 μg; Day 254; Test type: Superiority; p = 0.188, MMRM; LS Mean = 0.071, 95% CI 2-sided [-0.035 to 0.178], Standard Error of Mean 0.0542
Statistical Analysis 11: Comparison: QMF149 150/160 μg vs MF 400 μg; Day 254; Test type: Superiority; p = 0.002, MMRM; LS Mean = 0.168, 95% CI 2-sided [0.061 to 0.274], Standard Error of Mean 0.0543
Statistical Analysis 12: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Day 254; Test type: Superiority; p = 0.258, MMRM; LS Mean = 0.061, 95% CI 2-sided [-0.045 to 0.166], Standard Error of Mean 0.0538
Statistical Analysis 13: Comparison: QMF149 150/320 μg vs MF 800 μg; Day 364; Test type: Superiority; p = 0.154, MMRM; LS Mean = 0.079, 95% CI 2-sided [-0.030 to 0.187], Standard Error of Mean 0.0552
Statistical Analysis 14: Comparison: QMF149 150/160 μg vs MF 400 μg; Day 364; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.191, 95% CI 2-sided [0.082 to 0.299], Standard Error of Mean 0.0553
Statistical Analysis 15: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Day 364; Test type: Superiority; p = 0.455, MMRM; LS Mean = 0.041, 95% CI 2-sided [-0.067 to 0.148], Standard Error of Mean 0.0548

25. Secondary Outcome: Trough FEV1 Measured After 26 Weeks of Treatment
Description: as for outcome 1
Time Frame: Week 26
Population: FAS consisted of all participants in the RAN set who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | QMF149 150/320 μg | QMF149 150/160 μg | MF 800 μg | MF 400 μg | Salmeterol/Fluticasone 50/500 μg
Number analyzed (Participants) | 395 | 389 | 372 | 376 | 391
L | 2.383 (0.0159) | 2.387 (0.0160) | 2.250 (0.0162) | 2.176 (0.0162) | 2.346 (0.0160)
Statistical Analysis 1: Comparison: QMF149 150/320 μg vs Salmeterol/Fluticasone 50/500 μg; Test type: Non-Inferiority — QMF 150/320 was considered non-inferior to S/F 50/500 if the lower bound of the 95% CI was above the non-inferiority margin of -90 mL and was considered superior if the lower bound of the 95% CI was > 0. The p-value is for null-hypothesis testing; p = 0.101, MMRM; LS Mean = 0.036, 95% CI 2-sided [-0.007 to 0.080], Standard Error of Mean 0.0222

26. Secondary Outcome: Percentage of Participants With Composite Endpoint of Serious Asthma Outcomes
Description: A composite endpoint of serious asthma outcomes is defined as asthma-related hospitalization, asthma-related intubation, or asthma-related death and was reviewed by the Adjudication Committee.
Time Frame: Up to Week 52
Population: Safety Set consisted of all participants who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | QMF149 150/320 μg | QMF149 150/160 μg | MF 800 μg | MF 400 μg | Salmeterol/Fluticasone 50/500 μg
Number analyzed (Participants) | 443 | 437 | 440 | 443 | 444
percentage of participants | 0.7 | 0.5 | 1.6 | 1.8 | 0.5

27. Secondary Outcome: Percentage of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: An AE is any untoward medical occurrence (i.e., any unfavorable and unintended sign including abnormal laboratory findings, symptom or disease) in a participant or clinical investigation participant after providing written informed consent for participation in the study. An SAE is defined as any adverse event (appearance of (or worsening of any pre-existing) undesirable sign(s), symptom(s) or medical conditions(s) which meets any one of the following criteria: is fatal or life-threatening, results in persistent or significant disability/incapacity, constitutes a congenital anomaly/birth defect, requires inpatient hospitalization or prolongation of existing hospitalization or is medically significant, i.e. defined as an event that jeopardizes the participants or may require medical or surgical intervention.
Time Frame: Approximately up to 56 weeks
Population: Safety Set consisted of all participants who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | QMF149 150/320 μg | QMF149 150/160 μg | MF 800 μg | MF 400 μg | Salmeterol/Fluticasone 50/500 μg
Number analyzed (Participants) | 443 | 437 | 440 | 443 | 444
percentage of participants
  Adverse Events(AEs) | 64.6 | 66.8 | 70.0 | 72.2 | 65.3
  Serious Adverse Events(SAEs) | 4.7 | 4.6 | 4.8 | 7.0 | 4.7

ADVERSE EVENTS:
Time Frame: Serious adverse events: From first dose up to 30 days post last dose (approximately 56 weeks) Other adverse events: From first dose up to 7 days post last dose (approximately 53 weeks)
Description: The Safety Set consisted of all participants who received at least one dose of study medication.
Groups:
- QMF 150/320: QMF149 (Indacaterol acetate/Mometasone furoate) 150/320 μg was delivered o.d. via Concept1 inhaler in the evening.
- QMF 150/160: QMF149 (Indacaterol acetate/Mometasone furoate) 150/160 μg was delivered o.d. via Concept1 inhaler in the evening.
- MF 800: MF 800 μg of total daily dose (400 μg twice daily, in the morning and in the evening) was delivered via Twisthaler®.
- MF 400: MF 400 μg was delivered o.d. via Twisthaler® in the evening.
- S/F 50/500: Salmeterol xinafoate/fluticasone propionate 50/500 μg was delivered twice daily (in the morning and in the evening) via Accuhaler®.
Arm/Group | QMF 150/320 | QMF 150/160 | MF 800 | MF 400 | S/F 50/500
All-Cause Mortality (participants affected / at risk) | 0/443 | 0/437 | 0/440 | 1/443 | 0/444
Serious Adverse Events (participants affected / at risk) | 21/443 | 20/437 | 21/440 | 31/443 | 21/444
Other Adverse Events (participants affected / at risk) | 228/443 | 233/437 | 263/440 | 290/443 | 239/444
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QMF 150/320 (N=443) | QMF 150/160 (N=437) | MF 800 (N=440) | MF 400 (N=443) | S/F 50/500 (N=444)
Acute myocardial infarction (Cardiac disorders) | 2 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Goitre (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Corneal deposits (Eye disorders) | 0 | 1 | 0 | 0 | 0
Optic ischaemic neuropathy (Eye disorders) | 0 | 0 | 0 | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Complicated appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Dengue fever (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastroenteritis salmonella (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 1 | 0 | 3
Pneumonia (Infections and infestations) | 1 | 3 | 5 | 2 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sialoadenitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Accidental device ingestion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Eye injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Cerebellar haematoma (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Migraine with aura (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Vertebral artery aneurysm (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Calculus urethral (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Hydroureter (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Ureteric stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Cervix enlargement (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 6 | 8 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Chronic rhinosinusitis with nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Aortic dissection (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QMF 150/320 (N=443) | QMF 150/160 (N=437) | MF 800 (N=440) | MF 400 (N=443) | S/F 50/500 (N=444)
Diarrhoea (Gastrointestinal disorders) | 3 | 9 | 5 | 4 | 9
Bronchitis (Infections and infestations) | 20 | 22 | 22 | 21 | 17
Gastroenteritis (Infections and infestations) | 4 | 9 | 4 | 6 | 8
Influenza (Infections and infestations) | 12 | 13 | 19 | 10 | 15
Nasopharyngitis (Infections and infestations) | 50 | 58 | 78 | 82 | 47
Pharyngitis (Infections and infestations) | 10 | 11 | 12 | 12 | 14
Respiratory tract infection viral (Infections and infestations) | 10 | 16 | 14 | 12 | 13
Rhinitis (Infections and infestations) | 10 | 10 | 9 | 5 | 8
Upper respiratory tract infection (Infections and infestations) | 22 | 27 | 40 | 37 | 38
Upper respiratory tract infection bacterial (Infections and infestations) | 5 | 7 | 6 | 14 | 8
Viral infection (Infections and infestations) | 7 | 8 | 11 | 7 | 6
Viral upper respiratory tract infection (Infections and infestations) | 7 | 11 | 21 | 20 | 21
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 17 | 9 | 5 | 8
Headache (Nervous system disorders) | 26 | 21 | 24 | 23 | 22
Asthma (Respiratory, thoracic and mediastinal disorders) | 112 | 113 | 157 | 194 | 137
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 9 | 12 | 15 | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 | 6 | 8 | 9 | 8
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 5 | 11 | 7 | 11 | 7
Hypertension (Vascular disorders) | 10 | 14 | 13 | 11 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2018-01-17): https://cdn.clinicaltrials.gov/large-docs/86/NCT02554786/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-27): https://cdn.clinicaltrials.gov/large-docs/86/NCT02554786/SAP_001.pdf